

# Statistical Analysis Plan

Protocol Title A Phase 2b randomized, open-label, controlled, single center

study in Plasmodium falciparum-infected and uninfected adults age 18-55 years old in Kenya to evaluate the efficacy of the delayed, fractional dose RTS,S/AS01  $_{\rm E}$  malaria vaccine in subjects treated with artemisinin combination therapy plus

primaquine

**Protocol Number** CVIA 078, version 5.1, 24 May 2021

**Sponsor** PATH

**Principal Investigator** 

**Co-Principal Investigator** 

Version 4.0

**Date** Apr 15<sup>th</sup>, 2023

ClinicalTrials.gov NCT NCT04661579

Number

Version: 4.0  Date: Mar 5th, 2023

Protocol No. CVIA-078; RTS,S/AS01 E STATISTICAL ANALYSIS PLAN

# Statistical Analysis Plan (SAP) Approval Form

# PATH Reviewer Signature

This signature indicates approval for this SAP.

| Typed Name/Title | <u>Signature</u> | <u>Date</u> |
|--------------------|------------------|-------------|
| Statistician, PATH | | 14-Apr-2023 |

Author Signature

This signature indicates that appropriate and accurate information has been included in this SAP.

| Typed Name/Title | <u>Signature</u> | <u>Date</u> |
|---|---|---|
| Data Sciences Lead,<br>DF/Net Research, Inc. | | 14-Apr-2023 |

Version: 4.0 

# **Revision History**

| <u>Version</u> | <u>Date</u> | Summary of Revision |
|---|---|---|
| 0.1 | March 22, 2021 | Initial version |
| 0.2 | April 02, 2021 | Added Shells |
| 0.3 | April 16, 2021 | Clean version for ERC |
| 0.4 | May 3, 2021 | Updated shells |
| 1.0 | May 17, 2021 | Final version |
| 1.1 | May 18th 2021 | Small update to clarify the Total cohort for efficacy and ATP cohort for efficacy population definition |
| 2.0 | May 20 <sup>th</sup> 2022 | Updated the protocol version, Co-PI, and the values that define a positive result for Anti-CS results |
| 2.1 | Sep 27 <sup>th</sup> 2022 | Added a new section on the Timing of Analysis |
| 3.0 | Nov 2 <sup>nd</sup> 2022 | Finalized for signature |
| 3.1 | Jan 31st 2023 | Updated the start of at risk to 7 days after dose 3 instead of 14 days after dose 3. Updated the shells |
| 3.2 | Feb 28 <sup>th</sup> 2023 | Added survival curves for exploratory analysis and updated the list of TLF shells |
| 4.0 | Mar 5 <sup>th</sup> 2023 | Finalized for signature |
| | Apr 14 <sup>th</sup> 2023 | Updated the model for immunogenicity group comparisons and associated TLF shells |


# Table of Contents

| 1. | LI | ST O | F ABBREVIATIONS | . 11 |
|---|---|---|---|---|
| 2. | IN | TRO | DUCTION | . 13 |
| | 2.1 | Bac | ckground and rationale | 13 |
| | 2.2 | Stu | dy Objectives | . 13 |
| | 2.2 | 2.1 | Primary Objective | . 13 |
| | 2.2 | 2.2 | Secondary Objective | 13 |
| | 2.2 | 2.3 | Exploratory Objective | . 14 |
| | 2.3 | Stu | dy Design and Study Endpoints | . 14 |
| | 2.3 | 3.1 | Study Design | . 14 |
| | 2.3 | 3.2 | Study Endpoints | 15 |
| | 2.4 | Raı | ndomization and Treatment Assignment | . 17 |
| | 2.5 | Sar | nple Size and Power Considerations | . 18 |
| 3. | GI | ENEI | RAL CONSIDERATIONS FOR DATA ANALYSES | . 20 |
| | 3.1 | Sta | tistical Hypotheses | . 20 |
| | 3.2 | De | finition of Populations to be Analyzed (Analysis Datasets) | 20 |
| | 3.2 | 2.1 | Enrolled population | 20 |
| | 3.2 | 2.2 | Total vaccinated cohort (TVC) | 20 |
| | 3.2 | 2.3 | Safety analysis population | . 20 |
| | 3.2 | 2.4 | According to protocol (ATP) cohort for efficacy | 21 |
| | 3.2 | 2.5 | Total cohort for efficacy | 21 |
| | 3.2 | 2.6 | ATP cohort for immunogenicity | . 21 |
| | 3.3 | Tin | ne Window for Analysis | 21 |
| | 3.4 | Mis | ssing Data and Outliers | . 23 |
| | 3.4 | 1.1 | Missing Data | . 23 |
| | 3.4 | 1.2 | Outliers | . 23 |
| | 3.5 | Dat | ta Handling Conventions and Transformations | 23 |
| | 3.6 | | tistical Summaries, Confidence Intervals and P values | |
| | 3.7 | Mu | ltiple Comparisons/Multiplicity | . 24 |


| | 3.8 | Interim Analysis and Final Analysis | . 24 |
|---|---|---|---|
| | 3.9 | Statistical Software | . 24 |
| 4. | SU | BJECT DISPOSITION | . 25 |
| | 4.1 | Subject Enrollment | . 25 |
| | 4.2 | Disposition of Subjects | . 25 |
| | 4.3 | Eligibility Criteria | . 25 |
| 5. | SU | BJECT CHARACTERISTICS AND ADHERENCE | . 26 |
| | 5.1 | Baseline Demographics and Characteristics | . 26 |
| | 5.2 | Subject Characteristics at Each Visit | . 26 |
| | 5.3 | Visit and Vaccination Adherence, Sample Availability | . 26 |
| | 5.4 | Anti-Malarial Compliance | . 26 |
| | 5.5 | Protocol Deviations | . 26 |
| 6. | AN | ALYSIS OF THE PRIMARY EFFICACY ENDPOINT | . 27 |
| 7. | AN | ALYSIS OF THE SECONDARY ENDPOINT(S) | . 28 |
| | 7.1 | Secondary Efficacy | . 28 |
| | 7.2 | Immunogenicity | . 28 |
| | 7.3 | Safety Analyses | . 29 |
| | 7.3 | .1 Definition | . 29 |
| | 7.3 | .2 Analysis of Safety Endpoints | . 30 |
| 8. | EX | PLORATORY ANALYSES | . 32 |
| 9. | LIS | ST OF TABLES, LISTINGS AND FIGURES | . 33 |
| 10 | . 1 | TLF SHELLS | . 34 |
| 11 | . 1 | TIMING OF ANALYSIS | . 34 |
| D] | ЕМО | GRAPHICS TABLES | . 37 |
| | Table | 10.1.1: Enrollment Status by Group | . 37 |
| | Table | 10.1.2: Summary of eligibility criteria | . 38 |
| | | 10.1.3: Summary of Demographics by Treatment (TVC, total efficacy cohort and Per | |
| | | col Populations) | |
| | | 10.1.4: Summary of HLA Typing by Treatment (TVC Population) | |
| | Table | 10.1.5: Protocol Deviations | . 42 |


| Table 10.1.6: Medical History |
|---|
| Table 10.1.7: Vital Signs |
| Table 10.1.8: Physical Examination |
| Table 10.1.9: Prior Medications |
| Table 10.1.10: Concomitant Medications |
| Table 10.1.11: Vaccine Administration |
| Table 10.1.12: Anti-Malarial Compliance |
| TABLE 10.1.13.1: VISIT ATTENDANCE (EPOCH 1)50 |
| TABLE 10.1.13.2: VISIT ATTENDANCE (EPOCH 2) |
| TABLE 10.1.13.3: VISIT ATTENDANCE (EPOCH 3) |
| VACCINE EFFICACY TABLES53 |
| Table 10.2.1.1 and 2. Vaccine efficacy (Group 1 vs Group 4): First Infection Events (FIEs) of <i>P. falciparum</i> during the Active Detection of Infection period by HIV status and overall (ATP cohort for efficacy and Total cohort for efficacy) |
| Table 10.2.2.1 and 2 Vaccine efficacy (Group 2 vs Group 5): First Infection Events (FIEs) of P. falciparum during the Active Detection of Infection period by HIV status and overall (ATP cohort for efficacy and Total cohort for efficacy) |
| Table 10.2.3.1 and 2 Vaccine efficacy (Group 1 vs Group 2): First Infection Events (FIEs) of <i>P. falciparum</i> during the Active Detection of Infection period by HIV status and overall (ATP cohort for efficacy and Total cohort for efficacy) |
| Table 10.2.4.1 and 2 Vaccine efficacy (Group 4 vs Group 5): First Infection Events (FIEs) of <i>P. falciparum</i> during the Active Detection of Infection period by HIV status and overall (ATP cohort for efficacy and Total cohort for efficacy) |
| Table 10.2.5.1 and 2 Summary of subjects at risk, person-time, number of FIEs and incidence rate (ATP cohort for efficacy and Total cohort for efficacy) for Group 1 and 4 |
| Table 10.2.6.1 and 2 Summary of subjects at risk, person-time, number of FIEs and incidence rate (ATP cohort for efficacy and Total cohort for efficacy) for Group 2 and 5 |
| Table 10.2.7.1 and 2 Summary of median time to FIEs and hazards (ATP cohort for efficacy and Total cohort for efficacy) |
| IMMUNOGENICITY TABLES60 |
| Table 10.3.1.1 and 2: Number and Percentage of Subjects with anti-CS NANP Antibody Titer/Avidity Equal to or above Cut-off (seropositive) and GMTs (ATP cohort for immunogenicity and Total vaccinated cohort) |


| | Table 10.3.2.1 and 2: Number and Percentage of Subjects with Anti-CS C-term Antibody Titer/Avidity Equal to or above Cut-off and GMTs (ATP cohort for immunogenicity and Total cohort for efficacy) |
|---|---|
| | Table 10.3.3.1 and 2: Number and Percentage of Subjects with Anti-HBsAb Titer Equal to or above Cut-off and GMTs (ATP cohort for immunogenicity and Total vaccinated cohort) 61 |
| | Table 10.3.4.1 and 2: Geometric Fold Rise in Anti-CS NANP Antibody Titer at Each Post-Vaccination Timepoint Compared to Screening (ATP cohort for immunogenicity and Total vaccinated cohort) |
| | Table 10.3.5.1 and 2: Geometric Fold Rise in Anti-CS C-term Antibody Titer at Each Post-Vaccination Timepoint Compared to Screening (ATP cohort for immunogenicity and Total vaccinated cohort) |
| | Table 10.3.6.1 and 2: Geometric Fold Rise in Anti-HBsAb Titer at Each Post-Vaccination Timepoint Compared to Screening (ATP cohort for immunogenicity and Total vaccinated cohort) |
| S | AFETY TABLES63 |
| | Table 10.4.1.1: Overall Safety Profile by Treatment (Safety Population) |
| | Table 10.4.1.2: Frequency of Local Solicited Adverse Events by Treatment and Severity (Safety Population) |
| | Table 10.4.1.3: Frequency of Systemic Solicited Adverse Events by Treatment and Severity (Safety Population) |
| | Table 10.4.1.4: Summary of Unsolicited Adverse Events by Treatment (Safety Population) . 67 |
| | Table 10.4.1.5: Summary of Unsolicited Adverse Events by Treatment, Severity and Relationship to Study Treatment (Safety Population) |
| | Table 10.4.1.6: Summary of Serious Adverse Events by Treatment (Safety Population) 70 |
| | Table 10.4.1.7: Frequency of Local Solicited Adverse Events by Treatment, Injection Period, and Severity (Safety Population) |
| | Table 10.4.1.8: Frequency of Systemic Solicited Adverse Events by Treatment, Injection Period, and Severity (Safety Population) |
| | Table 10.4.1.9: Summary of Adverse Events of Special Interest by Treatment (Safety Population) |
| | Table 10.4.1.10: Summary of Adverse Events (Safety Population) |
| | Table 10.4.1.11: Summary of Recurrent Adverse Events (Safety Population) |
| | Table 10.4.1.12: Summary of Adverse Events that Persisted beyond 6 Days Post-IP Administration (Safety Population) |


| | Table 10.4.1.13: Exploration of Group Comparisons for Common Adverse Events (Safety Population) | 80 |
|---|---|---|
| | Table 10.4.1.14: Safety Lab Data out of Range (Safety Population) | 81 |
| | Table 10.4.1.15: Summary of Safety Lab Results (Safety Population) | 82 |
| | Table 10.4.1.16: Summary of Hemoglobinopathy Results (Safety Population) | 83 |
| | Table 10.4.1.17: Summary of Urine Pregnancy Test Results (Safety Population) | 84 |
| | Table 10.4.1.18: Summary of All Non-Serious Adverse Events by Treatment (Safety Population) | 85 |
| 1 | 2. DEMOGRAPHICS LISTINGS | 86 |
| | Listing 10.1.1: Protocol Deviations | 86 |
| | Listing 10.1.2: Enrollment Status, Demographics and Subject Disposition | 87 |
| | Listing 10.1.3: Eligibility Criteria Not Met | 88 |
| | Listing 10.1.4: Listing of All Eligibility Criteria | 89 |
| | Listing 10.1.5: Baseline Demographics | 90 |
| | Listing 10.1.6: HIV Status and HLA Typing | 91 |
| | Listing 10.1.7: Prior Medications | 92 |
| | Listing 10.1.8: Concomitant Medication | 93 |
| | Listing 10.1.9: Medical History | 94 |
| | Listing 10.1.10.1: Visit Attendance (Epoch 1) | 95 |
| | Listing 10.1.10.2: Visit Attendance (Epoch 2) | 96 |
| | Listing 10.1.10.3: Visit Attendance (Epoch 3) | 97 |
| | Listing 10.1.11: Vaccine administration | 98 |
| | Listing 10.1.12: Anti-Malarials | 99 |
| | Listing 10.1.13: Vital Signs | 100 |
| | Listing 10.1.14: Physical Examinations | 101 |
| 1 | 3. SAFETY LISTINGS | 102 |
| | Listing 10.2.1: Solicited Adverse Events (Safety Population) | 102 |
| | Listing 10.2.2: Unsolicited Adverse Events (Safety Population) | 103 |
| | Listing 10.2.3: Serious Adverse Events (Safety Population) | 104 |
| | Listing 10.2.4: Adverse Events of Special Interest (Safety Population) | 105 |


| Lis | ting 10.2.5: Safety Laboratory Results (Safety Population) | 106 |
|---|---|---|
| Lis | ting 10.2.6: Hemoglobinopathy Tests Results (Safety Population) | 107 |
| Lis | ting 10.2.7: Urine Pregnancy Tests for Female Subjects (Safety Population) | 108 |
| 14. | IMMUNOGENICITY LISTING | 109 |
| Lis | ting 10.3.1: Listing of Antibody Titers/Avidity | 109 |
| 15. | VACCINE EFFICACY LISTING | 110 |
| Lis | ting 10.4.1 Listing of First Infection Events (FIEs) | 110 |
| Lis | ting 10.4.2 Listing of Parasitemia Test Results (ADI) | 111 |
| 16. | DEMOGRAPHICS FIGURES | 112 |
| Fig | gure 10.1.1: CONSORT Diagram | 112 |
| 17. | VACCINE EFFICACY FIGURES | 114 |
| Fig | gure 10.2.1: Kaplan-Meier survival curve for FIEs in Groups 1 and 4. | 114 |
| _ | gure 10.2.2: Kaplan-Meier survival curve for FIEs in Groups 1 and 4 stratified by HIV tus. 115 | |
| Fig | gure 10.2.3: Kaplan-Meier survival curve for FIEs in Groups 2 and 5. | 116 |
| _ | gure 10.2.4: Kaplan-Meier survival curve for FIEs in Groups 2 and 5 stratified by HIV tus. 117 | |
| Fig | gure 10.2.5: Kaplan-Meier survival curve for FIEs in Groups 1 and 2 | 117 |
| Fig | gure 10.2.6: Kaplan-Meier survival curve for FIEs in Groups 4 and 5 | 117 |
| _ | gure 10.2.7: Scaled Schoenfeld residuals with 95% confidence interval versus time for coups 1 and 4 FIEs during the entire study period (ATP cohort for efficacy) | 118 |
| _ | gure 10.2.8: Scaled Schoenfeld residuals with 95% confidence interval versus time for oups 2 and 5 FIEs during the entire study period (ATP cohort for efficacy) | 119 |
| _ | gure 10.2.9: Scaled Schoenfeld residuals with 95% confidence interval versus time for coups 1 and 2 FIEs during the entire study period (ATP cohort for efficacy) | 119 |
| _ | gure 10.2.10: Scaled Schoenfeld residuals with 95% confidence interval versus time for pups 4 and 5 FIEs during the entire study period (ATP cohort for efficacy) | 119 |
| 18. | IMMUNOGENICITY FIGURES | 120 |
| _ | gure 10.3.1: Reverse Cumulative Distribution Curves for Anti-CS NANP Antibody Titer<br>ch Group (ATP cohort for immunogenicity) | |
| | gure 10.3.2: Reverse Cumulative Distribution Curves for Anti-CS C-term Antibody Tites ch Group (ATP cohort for immunogenicity) | |


# Protocol No. CVIA-078; RTS,S/AS01 $_{\rm E}$ STATISTICAL ANALYSIS PLAN


# 1. LIST OF ABBREVIATIONS

ADI Active Detection of infection

AE Adverse Event

AESI Adverse event of special interest
A/L Artemether/lumefantrine
ALT Alanine aminotransferase
ATP According to protocol

anti-HBs Antibody to hepatitis B surface antigen

AS01 GSK's proprietary adjuvant system containing QS21,

MPL, and liposomes

CBC Complete Blood Count

CDC Centers for Disease Control and Prevention

CI Confidence interval
CMI Cell-mediated immunity
CRF Case report form

ELISA Enzyme-linked immunosorbent assay

GCP Good Clinical Practice
GMFRs Geometric Mean Fold Rises
GMT Geometric Mean Titer
CS Circumsporozoite protein
DHA/Pip Dihydroartemisinin-piperaquine
ELISA Enzyme-linked immunosorbent assay

GMT Geometric Mean Titer

H<sub>0</sub> Null hypothesis

H<sub>1</sub> Alternative hypothesis

Hb Haemoglobin HBsAb Hepatitis B sur

HBsAb Hepatitis B surface antibody
HBsAg Hepatitis B surface antigen
HIV Human immunodeficiency virus
ICF Informed Consent Form

ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee

IgG Immunoglobulin G
IP Investigational Product
LD PQ Low dose primaquine

AESI Adverse Events of Special Interest
MMRM Mixed Model for Repeated Measures
MedDRA Medical Dictionary for Regulatory Activities

NIH National Institutes of Health P. falciparum Plasmodium falciparum

PBMCs Peripheral Blood Mononuclear Cells

PCR Polymerase chain reaction


# Protocol No. CVIA-078; RTS,S/AS01 $_{\rm E}$ STATISTICAL ANALYSIS PLAN

| PLT | Platelet |
|-------|-------------------------------------------------------|
| PT | Preferred Term |
| RTS,S | Protein comprising CS and hepatitis B surface antigen |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SOC | System Organ Class |
| TVC | Total vaccine cohort |
| VE | Vaccine efficacy |
| WBC | White blood count |
| WHO | World Health Organization |


#### 2. INTRODUCTION

The main goal of this study is to assess the efficacy of RTS,S/AS01<sub>E</sub>, a candidate vaccine against malaria caused by *Plasmodium falciparum*, in adults positive for *P. falciparum* by PCR at baseline, but have been treated with anti-malarial medications to clear the parasite before receiving multiple doses of the vaccine. The goal is to overcome the reduced vaccine efficacy (hypo-responsiveness to the vaccine) reported in actively or chronically infected adults.

### 2.1 Background and rationale

In previous clinical trials for the RTS,S/AS01<sub>E</sub> vaccine, it has been reported that the vaccine has been less effective in adults in endemic regions. Adults living in areas of moderate to high malaria transmission often have co-existing asymptomatic circulating blood stage *P. falciparum* parasites that results from multiple exposures to infective mosquito bites. This has been recognized as inducing a level of immunologic hypo-responsiveness that may impede the development of a protective immune response following immunization. We hypothesize that treatment of malaria infection in individuals prior to immunization with the RTS,S/AS01 vaccine will reset the immune response to the vaccine and result in an increased vaccine efficacy.

The rationale of the trial is to compare the vaccine efficacy of RTS,S/AS01<sub>E</sub> in two groups of adults who differ with the presence/absence of baseline PCR-positive parasitemia. Both groups receive the same anti-malarial treatment to clear parasites or to prevent infection (prophylaxis) prior to immunization. A rabies comparator vaccine (Abhayrab) is administered to two parallel groups to assess the absolute vaccine efficacy (VE) against *P. falciparum* parasitemia and to investigate whether sub-optimal immune responses in previously infected or concurrently infected adults is a general phenomenon independent of the vaccine antigen.

# 2.2 Study Objectives

# 2.2.1 Primary Objective

To evaluate the vaccine efficacy assessed by time to first *P. falciparum* infection in RTS,S/AS01<sub>E</sub> vaccinated adults who are positive for *P. falciparum* by PCR at baseline and treated to clear parasites compared to adults administered a comparator Rabies vaccine (Abhayrab) who are also positive for *P. falciparum* by PCR at baseline and treated to clear parasites.

# 2.2.2 Secondary Objective

#### **Efficacy**

The secondary efficacy objective is to assess vaccine efficacy by time to first *P. falciparum* infection by PCR in RTS,S/AS01<sub>E</sub> vaccinated adults who are negative for *P. falciparum* at baseline and are provided anti-malarial chemo-prophylaxis versus the vaccine efficacy against *P.* 


*falciparum* of a comparator rabies vaccine that are administered to adults who are also negative for *P. falciparum* at baseline and receive the same anti-malarial chemo-prophylaxis.

# Safety

There are several secondary safety objectives for the trial:

- To assess the safety of RTS,S/AS01<sub>E</sub> in terms of serious adverse events (SAEs) during the whole study period (from Dose 1 to study conclusion)
- To assess the safety and reactogenicity of RTS,S/AS01<sub>E</sub> in terms of solicited local and systemic adverse
  events within 7 days after each vaccination in the first 50 subjects in groups 1 and 2, and in all 35 subjects
  from Group 3.
- To assess the safety of RTS,S/AS01<sub>E</sub> in terms of unsolicited adverse events within 28 days after each vaccination

### **Immunogenicity**

The secondary immunogenicity objective is to assess the level & avidity of anticircumsporozoite (CS) antibody, and that of hepatitis B surface antibodies (HBsAb), for groups 1, 2 and 3.



# 2.3 Study Design and Study Endpoints

#### 2.3.1 Study Design

The five groups for this study are summarized in Table 1. The schedules for immunization and anti-malarial treatment are listed in Table 2.

Table 1. The five study groups and their descriptors (from protocol)

| Group | Vaccine | Sample<br>size | Baseline<br>Parasitemia | Anti-malarial<br>Rx | Anti-malarial Ro<br>rationale |
|---|---|---|---|---|---|
| Group 1 | RTS,S/AS01E | 164 | + | #11 | Clear parasites |
| Group 2 | RTS,S/AS01E | 128 | 171 | + | Prophylaxis |
| Group 3 | RTS,S/AS01E | 35 | + | 5 | 100 |
| Group 4 | Rabies | 164 | + | Ťa | Clear parasites |
| Group 5 | Rabies | 128 | (±) | ¥s | Prophylaxis |


Table 2. The schedule of immunization and anti-malarial treatment (from protocol).

| Group | Month - | Month 0 | 1-2 wks before | Month 1 | 1 wk before | Month 7 | Month |
|---|---|---|---|---|---|---|---|
| | 1 | (Vaccine 1) | Vx dose 2 | (Vaccine 2) | Vx dose 3 | (Vaccine 3) | 8 to 14 |
| Group 1 | DHA/Pip<br>+ LD PQ | RTS,S/AS01 <sub>E</sub> | DHA/Pip + LD<br>PQ | RTS,S/AS01 <sub>E</sub> | A/L + LD<br>PQ | 1/5 <sup>th</sup> dose<br>RTS,S/AS01 <sub>E</sub> | ADI |
| Group 2 | DHA/Pip<br>+ LD PQ | RTS,S/AS01 <sub>E</sub> | DHA/Pip + LD<br>PQ | RTS,S/AS01 <sub>E</sub> | A/L + LD<br>PQ | 1/5 <sup>th</sup> dose<br>RTS,S/AS01 <sub>E</sub> | ADI |
| Group 3 | - | RTS,S/AS01 <sub>E</sub> | - | RTS,S/AS01 <sub>E</sub> | - | 1/5 <sup>th</sup> dose<br>RTS,S/AS01 <sub>E</sub> | - |
| Group 4 | DHA/Pip<br>+ LD PQ | Rabies | DHA/Pip + LD<br>PQ | Rabies | A/L + LD<br>PQ | Rabies | ADI |
| Group 5 | DHA/Pip<br>+ LD PQ | Rabies | DHA/Pip + LD<br>PQ | Rabies | A/L + LD<br>PQ | Rabies | ADI |

**Group 1.** Subjects have detectable *P. falciparum* parasitemia at baseline measured by PCR. Anti-malarial treatment with DHA/Pip to clear asexual stage and young gametocyte parasites plus LD PQ to clear mature gametocytes will be given 4 weeks prior to immunization with RTS,S/AS01<sub>E</sub>. A 2<sup>nd</sup> course of DHA/Pip plus Primaquine will be given 2 weeks before second RTS,S/AS01<sub>E</sub> immunization. One week before 3<sup>rd</sup> RTS,S/AS01<sub>E</sub> immunization, a three-day course of A/L plus Primaquine will be administered to clear infection.

**Group 2.** Subjects have no detectable *P. falciparum* parasitemia as measured by PCR at enrolment. The same anti-malarial treatment regimen as for Group 1 will be administered before each dose of RTS,S/AS01<sub>E</sub> immunization as chemo-prophylaxis against *P. falciparum*.

**Group 3.** Subjects have detectable *P. falciparum* parasitemia at baseline measured by PCR but will not receive any anti-malarial medications to clear PCR-positive parasites. This group includes 35 subjects and is included only for immunological assessment and not for vaccine efficacy.

**Group 4.** Subjects have detectable *P. falciparum* parasitemia at baseline measured by PCR and will receive the same anti-malarial treatment on the same schedule as subjects in group 1. However, subjects in Group 4 will be administered the Abhayrab rabies vaccine instead of RTS,S/AS01<sub>E</sub>.

**Group 5.** Subjects have <u>no</u> detectable *P. falciparum* parasitemia as measured by PCR at enrolment and will receive the same anti-malarial treatment on the same schedule as subjects in group 2. Similarly, subjects in Group 5 will be administered the Abhayrab rabies vaccine instead of RTS,S/AS01 <sub>E</sub>.

# 2.3.2 Study Endpoints


Protocol No. CVIA-078; RTS,S/AS01 E STATISTICAL ANALYSIS PLAN

#### The primary endpoint

The primary endpoint is defined as the time to first PCR-detectable malaria infection in Groups 1 and 4 during the ADI phase of the study. Vaccine efficacy for subject in (Group 1) who are immunized with RTS,S/AS01 $_{\rm E}$  vaccine will be compared to volunteers in Group 4 who are immunization with a comparator rabies vaccine.

#### Secondary Endpoints

#### Secondary endpoint for vaccine efficacy:

The secondary endpoint is defined as the time to first PCR-detectable malaria infection in Groups 2 and 5 during the ADI phase of the study. Vaccine efficacy in group 2 subjects who are administered RTS, S/AS01  $_{\rm E}$  will be compared to volunteers in Group 5 who are immunized with a comparator rabies vaccine.

#### Secondary endpoint for safety:

- Frequency count and proportion of subjects reporting serious adverse events (SAEs) during the whole study
  period
- Frequency count and proportion of subjects reporting solicited local and systemic adverse events within 7 days after each vaccination
- Frequency count and proportion of subjects reporting unsolicited adverse events within 28 days after each
  vaccination

#### Secondary endpoint for immunogenicity:

- Anti-circumsporozoite (CS) antibody levels & avidity for subject in Groups 1,2 and 3.
- Hepatitis B surface antibody (HBsAb) levels for subjects in Groups 1,2 and 3.






# 2.4 Randomization and Treatment Assignment

This study is an open label study and eligible subjects will be stratified by baseline parasitemia status and block randomized. Among those positive for parasitemia at baseline a total of 363 will be randomized. The first 105 will be randomized in a 1:1:1 ratio with 35 subjects assigned to each of Groups 1, 3 and 4. The next 258 subjects with baseline parasitemia will be randomized in a 1:1 ratio to Groups 1 and 4 with a total of 129 additional subjects per group. Two hundred fifty-six subjects that are negative for parasitemia at baseline will be randomized with an 1:1 ratio to Groups 2 and 5. This randomization schedule will result in a total of 164, 128, 35, 164, and 128 for Groups 1 through 5, respectively (Table 1). In addition, HIV infection status will be noted prior to randomization, and individuals will be stratified across the groups to the extent possible. The proportion of subjects per group that are HIV positive rate for the groups will be capped near 20% for each group. The randomization scheme and the randomization lists with their block sizes used for the study is shown in Figure 1.




Figure 1. The schematic diagram of the randomization process for the study (from randomization plan). The HIV positive rate for each group are capped near 20%.

# 2.5 Sample Size and Power Considerations

This is a Phase 2b study to assess the vaccine efficacy of RTS,S/AS01  $_{\rm E}$  in adults in a malaria endemic region. The statistical analysis will measure vaccine efficacy using Cox proportional hazards regression model (time to first PCR-positive infection). An attack rate of 40% over 6 months has been assumed as a conservative estimate in an epidemiologic setting of perennial transmission in Western Kenya. A fixed vaccine efficacy of 50% is a conservative assumption according to the estimated vaccine efficacy.

Using an event-based design and assuming 10% drop out of the enrolled population and a one-sided  $\alpha$ =0.025, the following table lists the power and required number of events to conduct the analysis.


Table 3. Sample Size Calculations (from protocol)

| Power | N to enroll per group | Total events<br>required to<br>conduct<br>analysis | Endpoint |
|---|---|---|---|
| 90% | 164 | 92 | Primary (Group 1 vs 4) |
| 80% | 128 | 72 | Secondary (Group 2 vs 5) |

The impact of the event-driven design is that the study will continue to follow up until 92 first PCR-positive infection events, subsequently referred to as events, have been observed in aggregate between Groups 1 and 4, and 72 events have been observed in the aggregate of Groups 2 and 5. If the aggregate numbers of events have been reached prior to 24 weeks of ADI, study actives will continue to occur through the end of the ADI. If the aggregate number of events during ADI does not reach the cutoff indicated in Table 3, then the ADI will be extended up to 48 weeks or until the total number of events is reached, whichever occurs first. This will require the PCR lab to provide timely aggregated reports of event counts (across Group 1 plus 4; and Group 2 plus 5) and may result in more than the required events for either the primary or secondary endpoint.

An additional cross-sectional PCR will be performed at the Study Termination Visit, but these PCR results will not count toward the study endpoints.

Based on these assumptions we estimate a greater than 90% probability of observing the required number of events for the primary and secondary analyses by 6.9 months. However, larger dropout rates and/or a lower attack rate might extend the amount of follow-up time necessary to accumulate the required number of events.

The sample size for the immunologic sub-cohort (CMI assays in all subjects in RTS,S/AS01  $_{\rm E}$  groups 1, 2, and 3) is based on logistical considerations and the feasibility of the collection and processing of PBMCs. Analysis of these exploratory endpoints and inter-group differences will be descriptive in nature.


# 3. GENERAL CONSIDERATIONS FOR DATA ANALYSES

# 3.1 Statistical Hypotheses

The primary and secondary hypotheses will be assessed using Cox proportional hazards regression (time to first PCR-positive infection). These hypotheses tests will be supplemented with two-sided confidence intervals for the hazard ratios as described below.

The null  $(H_0)$  and alternative  $(H_1)$  hypotheses for the primary analysis of time to first malaria infection in Groups 1 and 4 is as follows:

H<sub>0</sub>: Among adults positive for *P. falciparum* at baseline the hazard rate for first malaria infection for RTS,S/AS01<sub>E</sub> vaccinated adults (Group 1) is not different than that of adults administered the comparator rabies vaccine (Group 4) as measured by the hazard ratio.

H<sub>1</sub>: Among adults positive for *P. falciparum* at baseline the hazard rate for malaria infection for RTS, S/AS01<sub>E</sub> vaccinated adults (Group 1) is different than that of adults administered the comparator rabies vaccine (Group 4) as measured by the hazard ratio.

The null and alternative hypotheses for the secondary efficacy analysis of time to first malaria infection in Groups 2 and 5 is as follows:

H<sub>0</sub>: Among adults negative for *P. falciparum* at baseline the hazard rate for malaria infection for RTS,S/AS01E vaccinated adults (Group 2) is not different than that of adults administered the comparator rabies vaccine (Group 5) as measured by the hazard ratio.

H<sub>1</sub>: Among adults negative for *P. falciparum* at baseline the hazard rate for first malaria infection for RTS,S/AS01<sub>E</sub> vaccinated adults (Group 2) is different than that of adults administered the comparator rabies vaccine (Group 5) as measured by the hazard ratio.

# 3.2 Definition of Populations to be Analyzed (Analysis Datasets) 3.2.1 Enrolled population

All subjects who have provided written informed consent, regardless of the subject's screening, randomization, and vaccination status in the study.

# 3.2.2 Total vaccinated cohort (TVC)

All subjects in the enrolled population who are randomized and received at least one vaccination.

# 3.2.3 Safety analysis population

All subjects in the TVC for which any safety data is available. All safety analyses will be performed using this population. The denominators for different safety endpoints may vary according to the number of subjects with available data for the specific endpoint.


#### 3.2.4 According to protocol (ATP) cohort for efficacy

The ATP cohort for efficacy will include all subjects included in the TVC with no major protocol deviations that are determined to potentially interfere with the efficacy assessment of the study vaccine and contributed to the time at risk starting 7 days after the third dose. The membership in this study population will be determined in a blinded fashion at a data review meeting attended by the sponsor Medical Officer, the site PI/Co-PI, and the sponsor Statistician. The list of criteria used to exclude subjects from ATP, including anti-malarial administration and other relevant analysis protocol deviations, will be finalized before database freeze. The details can be found in the Note to File (NTF) from the meeting.

# 3.2.5 Total cohort for efficacy

Given the potential for some participants to receive COVID-19 vaccine during the study, an additional total efficacy cohort is defined to include all TVC subjects who receive all three doses of RTS,S/AS01<sub>E</sub> vaccine or comparator and contribute to time at risk starting 7 days after the third dose.

#### 3.2.6 ATP cohort for immunogenicity

The ATP cohort for immunogenicity will include all subjects included in the TVC with no major protocol deviations that are determined to potentially interfere with the immunogenicity assessment of the study vaccine. This population will serve as the primary analysis population for the immunogenicity endpoints. The population will be adapted by time point to include all eligible subjects' data up to the time of disqualifying protocol deviation. The criteria used to exclude subjects from this cohort will include but not limited to: performed blood samplings for immunogenicity according to protocol intervals; did not use any medication or blood products forbidden by the protocol; did not have any reported underlying medical condition influencing immune responses. Similarly, the membership in this study population will be determined in a blinded fashion at a data review meeting attended by the sponsor, investigator, and DFnet and finalized before database freeze. The details can be found in the Note to File (NTF) from the meeting.

# 3.3 Time Window for Analysis

Study day will be calculated as the actual date minus date of the first dose of vaccine (Day 1) + 1 and will be used to show start/ stop day of assessments and events. If the event date is partial or missing, the corresponding study day and study duration will appear partial or missing in the listings.

Study day is defined to account for potential deviation from the visit schedule and unscheduled visits, all by-visit summary tables, unless otherwise specified, will be based on analysis visits, which will be assigned based on time window around the scheduled visit days below. However, listings will include all scheduled, unscheduled, retest and early withdrawal data. In general:


- unscheduled measurements will not be included if they do not fall within the analysis window listed below, but will contribute to the baseline value, or best/worst case value where required (e.g. shift table).
- for retest measurements (with same visit number assigned or fall within the same time window as another measurement), the last available measurement for that visit will be used with the exception for ADI visits where the first result will be used.
- early withdrawal data will be mapped to the next available visit number.

The following general time windows will be used:

Table 4. Time windows for Analysis

| Scheduled time point | Study Day Window |
|----------------------|------------------|
| Visit 2 | Day -29 to -25 |
| Visit 5 | Day -3 to 4 |
| Visit 7 | Day 8 to 10 |
| Visit 11 | Day 26 to 32 |
| Visit 12 | Day 36 to 38 |
| Visit 13 | Day 54 to 60 |
| Visit 14 | Day 188 to 192 |
| Visit 17 | Day 194 to 200 |
| Visit 18 | Day 204 to 206 |
| Visit 19 | Day 208 to 214 |
| Visit 20 | Day 221 to 229 |
| Visit 21 | Day 242 to 250 |
| Visit 22 | Day 263 to 271 |
| Visit 23 | Day 284 to 292 |
| Visit 24 | Day 305 to 313 |
| Visit 25 | Day 326 to 334 |
| Visit 26 | Day 347 to 355 |
| Visit 27 | Day 368 to 376 |
| Visit 28 | Day 389 to 397 |
| Visit 29 | Day 410 to 418 |
| Visit 30 | Day 431 to 439 |
| Visit 31 | Day 452 to 460 |
| Visit 32 | Day 473 to 481 |
| Visit 33 | Day494 to 502 |
| Visit 34 | Day 514 to 523 |
| Visit 35 | Day 536 to 544 |


# 3.4 Missing Data and Outliers

# 3.4.1 Missing Data

Non-missing ELISA data are considered validated. Missing ELISA data are considered non-retrievable. They will not be imputed and will be analyzed as if they were randomly missing. For subjects who discontinue from the study, their immunogenicity data collected before discontinuation will be analyzed under the analysis populations as applicable.

If severity or relationship to the IP administration for a reported AE or serious adverse event (SAE) is missing, an independent category "Missing" will be reported. If a start or stop date associated with a reported concomitant medication, AE, or SAE is incomplete or missing, the following rules will be applied:

- If the day of the start date is missing and the month and year of the start date are known, compare the start month and year to the month and year of visits 1 3. If the start month and year match exactly one of visits 1 3, then use the day of the date of that matched visit; otherwise use the 15th day of the month.
- · If either month or year is missing, no imputations will be done.

If stop date for a concomitant medication/medical history (AE or SAE) is missing, the medication/medical history will be considered ongoing.

If the study termination date is missing, it will not be imputed.

# 3.4.2 Outliers

Graphic inspection for outliers will be performed. No data will be excluded from the primary and secondary analyses, including any outliers. All transformations of the study data will be prespecified.

### 3.5 Data Handling Conventions and Transformations

The antibody titers will be transformed using log10 transformation for geometric mean analyses. Data will be back transformed to the original scale for presentation.

# 3.6 Statistical Summaries, Confidence Intervals and P values

Continuous data will be summarized by vaccination group with number of observations (n), mean, standard deviation (SD), median, Interquartile range, minimum, and maximum; Categorical results will be summarized by number of participants (n) and percentage (%) of subjects per vaccination group and visit. Unless otherwise specified, all statistical tests will be two-sided with a significance level of 0.05 and a 95% CI will be provided for estimates, as appropriate.


# 3.7 Multiple Comparisons/Multiplicity

No multiplicity adjustments will be performed.

# 3.8 Interim Analysis and Final Analysis

There is no planned interim analysis for the study.

A final analysis on all efficacy, safety and immunogenicity data will be performed after the study ends, when all additional safety data has been collected following the last subject's last study visit and the database is cleaned and locked.

#### 3.9 Statistical Software

All statistical analyses will be performed using SAS® software version 9.4 or later.


# 4. SUBJECT DISPOSITION

# 4.1 Subject Enrollment

Expected and actual subject enrollment will be tabulated by study group. The number and proportion of screened subjects meeting and not meeting entry criteria will also be tabulated.

# 4.2 Disposition of Subjects

Subject disposition will be summarized by study group. The following information will be tabulated. Summaries of subject disposition will be prepared for all subjects, including the number and percent enrolled, screened, randomized, and administered antimalarials and vaccines [T.10.1.1, L.10.1.2], as well as a CONSORT diagram [F.10.1.1] describing study participation and discontinuation. The reasons for screen failures, discontinuations, and population exclusions will be summarized and listed [T.10.1.5, L.10.1.1].

# 4.3 Eligibility Criteria

The inclusion and exclusion criteria used for screening in this study are listed in the protocol. The subjects excluded from the study for failing each inclusion/exclusion criteria and exclusion criteria will be listed and summarized [T.10. 1.2, L.10.1.3]


#### 5. SUBJECT CHARACTERISTICS AND ADHERENCE

#### 5.1 Baseline Demographics and Characteristics

Baseline demographics and characteristics, including age, height, weight, BMI, sex, race, and HIV status will be summarized for the TVC, total efficacy cohort and per protocol populations by vaccination group using descriptive statistics (mean, standard deviation, median, interquartile range, minimum and maximum for continuous features and rates for categorical features). [T.10.1.3, L.10.1.4]

Medical history will be tabulated by Medical Dictionary for Regulatory Activities (MedDRA v23) System Organ Class (SOC), Preferred Term (PT) and vaccination group. For the TVC population, medical history will be listed and summarized by category [T.10.1.6, L.10.1.9]. Using the World Health Organization (WHO, version: Mar2020) Drug Dictionary, prior and concomitant medications will be tabulated by anatomical therapeutic chemical (ATC) classification, preferred drug name and vaccination group [T.10.1.9, T.10.1.10, L.10.1.7, L.10.1.8].

#### 5.2 Subject Characteristics at Each Visit

Vital signs [T.10.1.7] and physical exam results [T.10.1.8] collected at other visits will be summarized for the TVC, total cohort for efficacy and per protocol populations by vaccination group.

Listings of vital signs [L.10.1.13] and physical exam results [L.10.1.14] at each applicable time point will be provided at participant-level.

#### 5.3 Visit and Vaccination Adherence, Sample Availability

A summary and listing of visit attendance [T.10.1.13.1-3, L.10.1.10.1-3] will be prepared, in addition to a summary and listing of vaccine administration and sample collection/availability for each sample [T.10.1.11, L.10.1.11].

#### 5.4 Anti-Malarial Compliance

The detailed information on the administration of three anti-malarials used in this study will be listed for the SAF population, including number of tablets dispensed, number of tablets returned, date, time, and compliance of dosing. Furthermore, since anti-malarial treatment does not allow for missed doses, their compliances will be listed by visits and summarized as the number and percentage of participants who have missed at least one dose of anti-malarials [T.10.1.12, L.10.1.12].

# 5.5 Protocol Deviations

A summary and listing of protocol deviations will be prepared [T.10.1.5, L.10.1.1].


Document ID: 2940b9f833d20dadf1251001aa420c67b5b7d78213e65c8226c47e70a74c3f5a

#### 6. ANALYSIS OF THE PRIMARY EFFICACY ENDPOINT

Vaccine efficacy against the first PCR-positive *P. falciparum* infection among adults who were *P. falciparum* positive at baseline will be assessed using Cox proportional hazards regression model with a covariate for group assignment to compare Groups 1 and 4. Specifically, the elapsed time starting 7 days after the third vaccination to the first PCR-positive *P. falciparum* detection or censoring will be analyzed. Time at risk will be presented as person years at risk (PYAR) dividing the days at risk by 365.25. As HIV status is a stratification factor in the randomization, it will be also included as covariate. An exploratory analysis, including Age, Gender and other baseline features might also be included as stratifications for the model if there is a randomization imbalance. Listing of FIEs and parasitemia testing results during ADI will be provided [L10.4.1 and L10.4.2].

The vaccine efficacy estimates (1-hazard ratio), 95% CI, and p-values will be calculated from this model using the Wald test. Ties will be handled using the Efron method [T.10.2.1]. In addition, tests and graphs based on the scaled Schoenfeld residuals will be used to assess the proportional hazard assumption [F10.2.5]. The interaction between HIV status and group assignment will be evaluated using a Wald test.

Descriptive statistics for each vaccination group and visit, the number of subjects at risk, persontime, number of PCR-confirmed first *P. falciparum* events and incidence rate will be tabulated [T.10.2.5]. The censoring rules are summarized in table 5. Similar tables will describe the median time-to-event and accumulative hazard from the cox regression model [T.10.2.7]. Survival curves for each vaccine group will be calculated non-parametrically, tabulated and presented graphically overall and by HIV status using the Kaplan-Meier method [F10.1.1-2].

This analysis will be conducted using both the ATP cohort for efficacy and the total cohort for efficacy.


#### 7. ANALYSIS OF THE SECONDARY ENDPOINT(S)

#### 7.1 Secondary Efficacy

Vaccine efficacy against the first PCR-positive *P. falciparum* infection among adults who were *P. falciparum* negative at baseline will be assessed using Cox proportional hazards regression with a covariate for group assignment to compare Groups 2 and 5. Similarly, HIV status, age, gender and other features might also be included as stratifications for the model. The vaccine efficacy estimates (1-hazard ratio), 95% CI, and p-values will be calculated from this model using the Wald test. Ties will be handled using the Efron method [T.10.2.2].

Table 5. Censoring rules

| Situation | Censoring Rules |
|---|---|
| The FIEs for Groups 1&4 and 2&5 reached in Epoch 2 | The entire period of epoch 2 (1st ADI period) |
| The FIEs for Groups 1&4 and 2&5 reached in Epoch 3 | The visit when the number of FIEs for both groups reached their targets during 2 <sup>nd</sup> ADI period |
| The FIEs for Groups 1&4 and 2&5 did not reach at the | The entire period of epoch 2 and 3 (1st and 2nd ADI |
| end of Epoch 3 | period) |
| Early withdrawal | The last visit available |
| Subjects treated with non-protocol anti-malarial during | The last visit before anti-malarials were administration |
| either ADI period | |

Similar descriptive statistics table as in the primary efficacy endpoint will be provided, as well as a table for median time to event and accumulative hazard and the Kaplan-Meier survival curves for each vaccination group overall and stratified by HIV status [T.10.2.6, T.10.2.7, F.10.2.3-4]. And this analysis will be conducted using both the ATP cohort for efficacy and the total cohort for efficacy.

#### 7.2 Immunogenicity

There are two antibodies, anti-CS, an antibody against both central repeat region (NANP) and C-terminal region of circumsporozoite protein, and anti-HBs (against hepatitis B surface protein), will be included in antibody response analysis of secondary immunogenicity endpoints for Groups 1-3 (Table 6). The antibody titer and avidity against the NANP or C-terminal of CS protein will be analyzed for visits 2, 5, 11, 13, 17, 20, 27 and 35. Anti-HBs antibody titer will be analyzed for visits 2, 5, 11 and 20. The analysis will be based on the ATP for immunogenicity cohort unless a significant number of subjects have missing data (>10%), then a secondary analysis based on the TVC will be performed to complement the ATP analysis. For estimation of the geometric mean titer (GMT), geometric mean ratio (fold increases), and corresponding confidence limits, analyses will incorporate censoring where appropriate and log-scale coefficients will be back-transformed in order to compute the estimate and corresponding confidence limits for the relevant quantity.

To calculate the fold increases in the antibody titer, an ELISA titer for a given sample being tested for anti-CS antibody levels will be considered seropositive if its value is greater than the following Lower Limit of Quantifications (LLOQs): anti-CS NANP (1XPBS) 54.1 1/DIL, anti-CS NANP (4M UREA) 37.9 1/DIL, anti-CS C-Term (1XPBS) 89.4 1/DIL, anti-CS C-term (4M UREA) 37.5 1/DIL. ELISA titers for the anti-HBs antibody will be considered positive if its value is greater than 10 mIU/mL. Samples that do not generate above or equal to the cut-offs will be reported as LLOQ for analysis purposes. Geometric Mean Fold Rises (GMFRs) will be computed using standard two-sample methods for the log difference of the within-subject increase from baseline, with corresponding CIs computed via *t*-distribution, utilizing the antilog transformation to present the ratio. Analyses of binary variables will include 95% CIs computed via the Clopper-Pearson method, and antibody response rates between each other among Groups 1-3 will be compared using either Fisher's exact test or Chi-square test. Furthermore, at each visit, GMT will be compared among groups 1, 2 and 3 by a mixed model for repeated measures with the log-transformed antibody titer as dependent variable, groups, HIV status and their interaction term as covariates and subject as a random effect. Compound symmetry will be


assumed for the covariance structure. The comparison of the ratios of GMT (estimated treatment differences between groups at all post baseline visits) will be estimated from a similar mixed model for repeated measures.

Table 6. Sampling Visits for Immunogenicity Assessment (from Appendix F of protocol)

| SAMPLES<br>COLLECTED FOR | Visit # | 2 | 5 | 6 | 7 | 11 | 13 | 17 | 20 | 27 | Termination<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|
| IMMUNOGENICITY | Study day | -27 | 1 | 2 | 8 | 29 | 57 | 197 | 225 | 372 | TBD* |
| Secondary endpoint -<br>Groups 1, 2, 3 | | | | | | | | | | | |
| Groups 1, 2, 3 | anti-CS NANP<br>levels<br>anti-CS NANP<br>avidity<br>anti-CS C-term | • | | | | | | • | | | • |
| Serum | levels | • | • | | | | • | • | • | • | • |
| | anti-CS C-term<br>avidity<br>anti-HbsAb | • | • | | | • | • | • | • | • | • |
| | antibodies | • | • | | | • | | | • | | |

The number and proportion of subjects exhibiting positive responses and their GMTs will be assessed for each antigen (anti-CS NANP or anti-CS C-term) and conditions (1XPBS or 4M Urea), including the number and proportion exhibiting a seroresponse (defined as a positive response among subjects negative at baseline) [T.10.3.1-3]. Individual fold increases will be listed and summarized as GMFRs by vaccination groups and visits. Subjects showing  $\geq 2,3$  and 4-fold rises in their antibody titers will also be listed individually by visits and summarized by vaccination groups and visits [T.10.3.4-6]. Additionally, the distribution of antibody titers against three antigens will be summarized using reverse cumulative distribution curves [F.10.3.1-3]. A listing of titer values will also be included [L.10.3.1].

# 7.3 Safety Analyses7.3.1 Definition

# Solicited Adverse Event

**Solicited AEs** are pre-specified local and systemic AEs that occur relatively more frequently or are known to be associated with immunization, which are monitored actively as potential indicators of vaccine reactogenicity. The following specific solicited local and systemic AEs and their intensity scales will be monitored for this study and listed in Table 7:

Table 7. Intensity Scales for Solicited Symptoms in Adults

| • | | • |
|---|---|---|
| Pain at injection site | 0 | Absent |
| | 1 | Painful on touch |
| | 2 | Painful when limb is moved |
| | 3 | Pain that prevents normal activity |
| Swelling at injection site | 0 | Absent |
| | 1 | Present and is easily tolerated |
| | 2 | Present and interferes with normal activity |
| | 3 | Present and prevents normal activity |
| Fever | 0 | <37.5°C (99.5°F) |
| | 1 | 37.5°C (99.5°F) to 38.0°C (100.4°F) |
| | 2 | >38.0°C (>100.4°F) to 39.0°C (102.1°F) |
| | 3 | >39.0°C (102.1°F) |
| Headache | 0 | Normal |
| | 1 | Headache feeling is easily tolerated |
| | 2 | Headache feeling interferes with normal activity |
| | 3 | Headache feeling prevents normal activity |
| | 0 | Gastrointestinal symptoms normal |
| | 1 | Gastrointestinal symptoms that are easily tolerated |
| | 2 | Gastrointestinal symptoms that interfere with normal activity |


| Gastrointestinal symptoms | 3 | Gastrointestinal symptoms that prevent normal activity |
|---|---|---|
| Fatigue | 0 | Normal |
| | 1 | Fatigue that is easily tolerated |
| | 2 | Fatigue that interferes with normal activity |
| | 3 | Fatigue that prevents normal activity |
| Muscle ache | 0 | Absent |
| | 1 | Muscle ache that is easily tolerated |
| | 2 | Muscle ache that interferes with normal activity |
| | 3 | Muscle ache that prevents normal activity |

#### **Unsolicited Adverse Events**

Unsolicited AEs are any AEs reported spontaneously by the subject, observed by the study staff during study visits or those identified during review of medical records or source documents. Solicited AEs with an onset after the seven-day solicitation period will be considered unsolicited AEs. In the absence of a diagnosis, abnormal physical examination findings or abnormal clinical safety laboratory test results that are assessed by the investigator to be clinically significant will be recorded as an AE.

#### Adverse Events of Special Interest

AESIs are unsolicited AEs of specific interest for safety monitoring include all seizures occurring within 30 days post-vaccination, meningitis and potential immune-mediated diseases (pIMDs). The full list of pIMDs can be found in the protocol.

#### Serious Adverse Event

An SAE is any AE that results in any of the following outcomes:

- Death
- Is life-threatening (i.e., the subject was, in the opinion of the investigator, at risk of death at the time of the
  event; it does not refer to an event which hypothetically might have caused death if it were more severe)
- Requires inpatient hospitalization or prolongation of existing hospitalization
- Results in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- Congenital anomaly or birth defect
- Important medical event that may not result in one of the above outcomes but may jeopardize the health of
  the study subject or may require medical or surgical intervention to prevent one of the outcomes listed
  above.

#### 7.3.2 Analysis of Safety Endpoints

All safety assessments will take place using the safety analysis population, according to the vaccination groups. All subject-based percentages (solicited/unsolicited AEs, clinical safety laboratory abnormalities, etc.) will be supplemented with two-sided 95% CIs computed via the Clopper-Pearson method. Individual summaries (denominators for percentages) will be limited to the number of subjects within the appropriate analysis population with data available for analysis for the given endpoint. When an AE occurs more than once for a subject, the subject will be only counted once for the corresponding PT according to the maximum severity of the events.

The overall safety profile for overall and each group will be summarized by the number of all solicited adverse events, the frequencies of local and systemic adverse events among them, the number of unsolicited events, the number and the percentages of subjects with any unsolicited adverse events, the number of adverse events of special interest, the number and the percentages of subjects with any adverse events of special interest, the number of adverse events, the number and the percentages of subjects with any adverse events [T.10.4.1.1].

All solicited AEs will be summarized according to defined severity grading scales. Frequencies and percentages of subjects experiencing each solicited AE will be presented for each symptom severity [T.10.4.1.2-3, T.10.4.1.7-8]. Summary tables showing the occurrence of any local or systemic solicited AE overall and solicited AEs that persist up to 7 days post-administration of IP overall will also be presented [T.10.4.1.12]. Data listings of all solicited AEs will be provided


by subject [L.10.2.1]. For common AEs group comparisons, including each preferred terms, frequency of signs and symptoms and the occurrences of Grade 4 solicited and unsolicited general reactions, will be explored and tested using Fisher's exact test [T.10.4.1.13]. In addition to safety population, these analyses will be also performed using the TVC analysis population.

All unsolicited AEs with onset occurring up to 28 days after each vaccine dose will be assessed as either related or not related to IP by the investigator and will be recorded. Additionally, all AESIs/SAEs throughout the study will be summarized [T.10.4.1.6, T10.4.1.9]. The original verbatim terms used by investigators to identify AEs in the eCRFs will be mapped to PTs using MedDRA. The AEs will then be grouped by MedDRA PTs into frequency tables according to SOC. All reported AEs, as well as AEs assessed by the investigator as related to IP, will be summarized according to SOC, PT within SOC, and severity [T.10.4.1.4-5]. Data listings sorted by subject will be provided [L.10.2.2].

A summary table [T.10.4.1.10] will be prepared for unsolicited AEs comprised of the following categories:

- Unsolicited AEs
- Related unsolicited AEs
- AESIs
- Related AESIs
- SAEs
- Related SAEs
- SAEs leading to death
- Unsolicited AEs leading to subject discontinuation

An additional summary table will be provided including all AEs excluding SAEs, i.e., all solicited, unsolicited, and AESIs [T.10.3.1.18]. A descriptive summary of recurrent AEs [T.14.3.1.11] will also be generated. Listings of AESIs and SAEs sorted by subject will also be provided [L.10.2.3-4]

For clinical safety laboratory data collected on the same day of the first dose of vaccination, individual hemoglobin, WBC count, platelet count, ALT, and creatinine values will be presented as number of subjects out of range (above and below normal range as appropriate) and tabulated by study group [T.10.4.1.14]. In addition, summary statistics of the lab result values will be presented, including mean, standard deviation (SD), 95% CIs, median, and interquartile range [T.10.4.1.15]. A listing of lab results will also be included [L.10.2.5].

Hemoglobinopathy test result at screening and urine pregnancy test results at screening, Visit 2, 5, 8 and 17, will also be listed [L.10.2.6-7] and summarized by overall and each group [T.10.4.1.16-17].




Protocol No. CVIA-078; RTS,S/AS01  $_{\rm E}$   $\,$  STATISTICAL ANALYSIS PLAN  $\,$ 

Date: Mar 5th, 2023

# 9. LIST OF TABLES, LISTINGS AND FIGURES

| 70 1.1 1.0 1.1 | E H (0) 1 C |
|---|---|
| Table 10.1.1<br>Table 10.1.2 | Enrollment Status by Group Summary of eligibility criteria |
| Table 10.1.2 | Summary of Demographics by Treatment (TVC, total cohort for efficacy and Per |
| 14016 10.1.5 | Protocol Population) |
| Table 10.1.4 | Summary of HIV Status and HLA Typing by Treatment (TVC, total cohort for efficacy |
| | and Per Protocol Population) |
| Table 10.1.5 | Protocol Deviations |
| Table 10.1.6 | Medical History |
| Table 10.1.7 | Vital Signs |
| Table 10.1.8 | Physical Examination |
| Table 10.1.9 | Prior Medications |
| Table 10.1.10 | Concomitant Medications |
| Table 10.1.11 | Vaccine Administration |
| Table 10.1.12<br>Table 10.1.13.1 | Anti-Malarial Compliance Visit Attendance (Epoch 1) |
| Table 10.1.13.1 | Visit Attendance (Epoch 1) Visit Attendance (Epoch 2) |
| Table 10.1.13.2 | Visit Attendance (Epoch 2) Visit Attendance (Epoch 3) |
| Table 10.2.1.1 and 2 | Vaccine efficacy (Group 1 vs Group 4): First Infection Events (FIEs) of P. falciparum |
| | during the Active Detection of Infection period by HIV status and overall (ATP cohort |
| | for efficacy and total cohort for efficacy) |
| Table 10.2.2.1 and 2 | Vaccine efficacy (Group 2 vs Group 5): First Infection Events (FIEs) of P. falciparum |
| | during the Active Detection of Infection period by HIV status and overall (ATP cohort |
| | for efficacy and total cohort for efficacy) |
| Table 10.2.3.1 and 2 | Vaccine efficacy (Group 1 vs Group 2): First Infection Events (FIEs) of P. falciparum |
| | during the Active Detection of Infection period by HIV status and overall (ATP cohort<br>for efficacy and total cohort for efficacy) |
| Table 10.2.4.1 and 2 | Vaccine efficacy (Group 4 vs Group 5): First Infection Events (FIEs) of P. falciparum |
| 1 aoic 10.2.4.1 and 2 | during the Active Detection of Infection period by HIV status and overall (ATP cohort |
| | for efficacy and total cohort for efficacy) |
| Table 10.2.5.1 and 2 | Summary of subjects at risk, person-time, number of FIEs and incidence rate (ATP |
| | cohort for efficacy and total cohort for efficacy) for Group 1 and 4 |
| Table 10.2.6.1 and 2 | Summary of subjects at risk, person-time, number of FIEs and incidence rate (ATP |
| Table 10.2.7.1 and 2 | cohort for efficacy and total cohort for efficacy) for Group 2 and 5 |
| Table 10.2.7.1 and 2 | Summary of median time to FIEs and hazard rates (ATP cohort for efficacy and total cohort for efficacy) |
| Table 10.3.1.1 and 2 | Number and Percentage of Subjects with anti-CS NANP Antibody Titer/Avidity Equal |
| Table 10.5.1.1 and 2 | to or above Cut-off (seropositive) and GMTs (ATP cohort for immunogenicity and |
| | Total vaccinated cohort) |
| Table 10.3.2.1 and 2 | Number and Percentage of Subjects with Anti-CS C-term Antibody Titer/Avidity Equal |
| | to or above Cut-off and GMTs (ATP cohort for immunogenicity and Total vaccinated |
| T 11 10 2 2 1 1 2 | cohort) |
| Table 10.3.3.1 and 2 | Number and Percentage of Subjects with Anti-HBsAb Titer Equal to or above Cut-off and GMTs (ATP cohort for immunogenicity and Total vaccinated cohort) |
| Table 10.3.4.1 and 2 | Geometric Fold Rise in Anti-CS NANP Antibody Titer at Each Post-Vaccination |
| 1 abic 10.5.4.1 and 2 | Timepoint Compared to Screening (ATP cohort for immunogenicity and Total |
| | vaccinated cohort) |
| Table 10.3.5.1 and 2 | Geometric Fold Rise in Anti-CS C-term Antibody Titer at Each Post-Vaccination |
| | Timepoint Compared to Screening (ATP cohort for immunogenicity and Total |
| m.11.40.2 | vaccinated cohort) |
| Table 10.3.6.1 and 2 | Geometric Fold Rise in Anti-HBsAb Titer at Each Post-Vaccination Timepoint |
| Table 10.4.1.1 | Compared to Screening (ATP cohort for immunogenicity and Total vaccinated cohort) Overall Safety Profile by Treatment (Safety Population) |
| Table 10.4.1.1 | Frequency of Local Solicited Adverse Events by Treatment and Severity (Safety |
| 14010 10.7.1.2 | Population) |
| Table 10.4.1.3 | Frequency of Systemic Solicited Adverse Events by Treatment and Severity (Safety |
| | Population) |
| Table 10.4.1.4 | Summary of Unsolicited Adverse Events by Treatment (Safety Population) |
| Table 10.4.1.5 | Summary of Unsolicited Adverse Events by Treatment, Severity and Relationship to |
| T.11. 10.4.1.6 | Study Treatment (Safety Population) |
| Table 10.4.1.6<br>Table 10.4.1.7 | Summary of Serious Adverse Events by Treatment (Safety Population) Frequency of Local Solicited Adverse Events by Treatment, Injection Period, and |
| 1 4010 10.4.1./ | Severity (Safety Population) |
| Table 10.4.1.8 | Frequency of Systemic Solicited Adverse Events by Treatment, Injection Period, and |
| 14010 10.4.1.0 | Severity (Safety Population) |
| Table 10.4.1.9 | Summary of Adverse Events of Special Interest by Treatment (Safety Population) |
| Table 10.4.1.10 | Summary of Adverse Events (Safety Population) |
| Table 10.4.1.11 | Summary of Recurrent Adverse Events (Safety Population) |
| Table 10.4.1.12 | Summary of Adverse Events that Persisted beyond 6 Days Post-IP Administration |
| | (Safety Population) 47 |


| m 11 40 44 40 | In the second se |
|---|---|
| Table 10.4.1.13 | Exploration of Group Comparisons for Common Adverse Events (Safety Population) |
| Table 10.4.1.14 | Safety Lab Data out of Range (Safety Population) |
| Table 10.4.1.15 | Summary of Safety Lab Results (Safety Population) |
| Table 10.4.1.16 | Summary of Hemoglobinopathy Results (Safety Population) |
| Table 10.4.1.17 | Summary of Urine Pregnancy Test Results (Safety Population) |
| Table 10.4.1.18 | Summary of All Non-Serious Adverse Events by Treatment (Safety Population) |
| Listing 10.1.1 | Protocol Deviations |
| Listing 10.1.2 | Enrollment Status, Demographics and Subject Disposition |
| Listing 10.1.3 | Eligibility Criteria Not Met |
| Listing 10.1.4 | Listing of All Eligibility Criteria |
| Listing 10.1.5 | Baseline Demographics |
| Listing 10.1.6 | HIV Status and HLA Typing |
| Listing 10.1.7 | Prior Medications |
| Listing 10.1.8 | Concomitant Medication |
| Listing 10.1.9 | Medical History |
| Listing 10.1.10.1 | Visit Attendance (Epoch 1) |
| Listing 10.1.10.2 | Visit Attendance (Epoch 2) |
| Listing 10.1.10.3 | Visit Attendance (Epoch 3) |
| Listing 10.1.11 | Vaccine administration |
| Listing 10.1.12 | Anti-Malarials |
| Listing 10.1.13 | Vital Signs |
| Listing 10.1.14 | Physical Examinations |
| Listing 10.2.1 | Solicited Adverse Events (Safety Population) |
| Listing 10.2.2 | Unsolicited Adverse Events (Safety Population) |
| Listing 10.2.3 | Serious Adverse Events (Safety Population) |
| Listing 10.2.4 | Adverse Events of Special Interest (Safety Population) |
| Listing 10.2.5 | Safety Laboratory Results (Safety Population) |
| Listing 10.2.6 | Hemoglobinopathy Tests Results (Safety Population) |
| Listing 10.2.7 | Urine Pregnancy Tests for Female Subjects (Safety Population) |
| Listing 10.3.1 | Listing of Antibody Titers/Avidity |
| Listing 10.4.1 | Listing of FIEs |
| Listing 10.4.2 | Listing of Parasitemia Test Results |
| Figure 10.1.1 | CONSORT Diagram |
| Figure 10.2.1 | Kaplan-Meier survival curve for FIEs in Groups 1 and 4. |
| Figure 10.2.2 | Kaplan-Meier survival curve for FIEs in Groups 1 and 4 stratified by HIV status. |
| Figure 10.2.3 | Kaplan-Meier survival curve for FIEs in Groups 2 and 5. |
| Figure 10.2.4 | Kaplan-Meier survival curve for FIEs in Groups 2 and 5 stratified by HIV status. |
| Figure 10.2.5 | Kaplan-Meier survival curve for FIEs in Groups 1 and 2. |
| Figure 10.2.6 | Kaplan-Meier survival curve for FIEs in Groups 4 and 5. |
| Figure 10.2.7 | Scaled Schoenfeld residuals with 95% confidence interval versus time for Groups 1 and |
| - | 4 FIEs during the entire study period (ATP cohort for efficacy) |
| Figure 10.2.8 | Scaled Schoenfeld residuals with 95% confidence interval versus time for Groups 2 and |
| | 5 FIEs during the entire study period (ATP cohort for efficacy) |
| Figure 10.2.10 | Scaled Schoenfeld residuals with 95% confidence interval versus time for Groups 1 and |
| | 2 FIEs during the entire study period (ATP cohort for efficacy) |
| Figure 10.2.11 | Scaled Schoenfeld residuals with 95% confidence interval versus time for Groups 4 and |
| | 5 FIEs during the entire study period (ATP cohort for efficacy) |
| Figure 10.3.1 | Reverse Cumulative Distribution Curves for Anti-CS NANP Antibody Titers in Each |
| | Group (ATP cohort for immunogenicity) |
| Figure 10.3.2 | Reverse Cumulative Distribution Curves for Anti-CS C-term Antibody Titers in Each |
| | Group (ATP cohort for immunogenicity) |
| Figure 10.3.3 | Reverse Cumulative Distribution Curves for Anti-HBsAb Titers in Each Group (ATP |
| | cohort for immunogenicity) |

# 10. TLF SHELLS

The TLF shells are included in a separate document/attached in the end.

# 11. TIMING OF ANALYSIS

Upon completion of last visit for the final participant and availability of immunogenicity results, a partial lock of the database will be realized, and a topline analysis will be initiated to include the results for safety, efficacy and immunogenicity. Immunogenicity results will include the data available before the partial lock. Upon collection of the remainder of the data for immunogenicity and final database lock, the final analysis on immunogenicity will be performed.


# TFL Shells for Protocol CVIA 078; RTS,S/AS10 $_{\text{E}}$ corresponding to SAP v3.1

Protocol title: A Phase 2b randomized, open-label, controlled, single center study in Plasmodium falciparum-infected and uninfected adults age 18-55 years old in Kenya to evaluate the efficacy of the delayed, fractional dose RTS,S/AS01  $_{\rm E}$  malaria vaccine in subjects treated with artemisinin combination therapy plus primaquine

**Date created**: v0.1 April 06<sup>th</sup>, 2021 **Updated**: v0.3 April 16<sup>th</sup>, **2021**, **Updated**: v0.4, May 3<sup>rd</sup>, 2021,

Updated: v1.0/v1.1 May 17-18<sup>th</sup>, 2021 added Total cohort for efficacy population for efficacy

summary tables and Total vaccinated cohort for immunogenicity summary tables

 $\label{thm:continuous} \begin{tabular}{ll} $U$ pdated: Jan $31^{st}$, 2023, removed change from baseline and toxicity grades from safety lab summaries and listings; updated TLF headers and footers $$I$ is the continuous continuou$ 

**Updated:** Feb  $28^{th}$ , 2023, added two efficacy tables (Groups 1 vs 2 and 4 vs 5), four survival curves (groups 1 vs 2 and groups 4 vs 5), two residual plots and two efficacy listings (FIEs and parasitemia test results)

Updated: Mar  $5^{th}$ , 2023, finalized to v4.0 for signature and updated again on April  $14^{th}$ , updated the model for the pairwise comparisons of immunogenicity and the TLF shells associated with.


Document ID: 2940b9f833d20dadf1251001aa420c67b5b7d78213e65c8226c47e70a74c3f5a

Protocol No. CVIA-078; RTS,S/AS01  $_{\rm E}$  STATISTICAL ANALYSIS PLAN

### **DEMOGRAPHICS TABLES**

Table 10.1.1: Enrollment Status by Group

| Table 10.1.1: Enrollment Status by Group | | | | | | |
|---|---|---|---|---|---|---|
| • | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total |
| | (N=) | (N=) | (N = | (N=) | (N=) | (N=) |
| Informed Consent signed | | | | | | XXXX |
| Eligible | | | | | | XXXX |
| Randomized | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| Randomized but received no study product at D1 | xx | XX | XX | X | xx | X |
| Received study product at D1 | xx | xx | XX | X | xx | X |
| Subjects who completed study | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Received study product at D1 who discontinued early | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Event | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Death | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Lost to follow-up | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Physician decision | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Eligibility criteria not met | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Withdrawal by subject | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Study terminated by sponsor | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Protocol deviation | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Other | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total vaccinated cohort, | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Safety analysis population, | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATP for efficacy | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATP for immunogenicity | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Total cohort for efficacy | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) |
| Total cohort for immunogenicty | (%X.XX) XX | (%X.XX) XX | (%X'XX) XX | (%X:XX) XX | (%X.XX) XX | (%x.xx) xx |

Total cohort for immunogenic,y
N: Number of subjects in each group.
Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 4: Rabies with anti-malarials to prevent infection (prophylaxis).
Denominator of percentage is number of subjects randomized and received at least one dose of IP.

 Date: Mar 5th, 2023 Version: 4.0

# Protocol No. CVIA-078; RTS,S/AS01<sub>E</sub> STATISTICAL ANALYSIS PLAN

| rable 10.1.2: Summary of engionity effects | Total<br>n (%) |
|---|---|
| Informed Consent Signed | XXXX |
| Subjects who met all eligibility criteria | xx (xx.x%) |
| Subjects who did not satisfy at least one eligibility criterion | xx (xx.x%) |
| Subjects who did not meet at least one Inclusion Criterion | xx (xx.x%) |
| Subject has provided signed or thumb printed and dated informed consent form | xx (xx.x%) |
| Subject has stated willingness to comply with all study procedures and availability for the duration of the study. | xx (xx.x%) |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xx (xx.x%) |
| Subjects who met at least one Exclusion Criterion | xx (xx.x%) |
| Subject has planned administration/administration of a vaccine not foreseen by the study protocol from within 30 days before the first dose of study vaccine until 30 days after the last dose of study vaccine | xx (xx.x%) |
| Subject has prior receipt of any rabies vaccine or experimental malaria vaccine. | xx (xx.x%) |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | xx (xx.x%) |
| | xx (xx.x%) |
| | xx (xx.x%) |
| | xx (xx.x%) |
| | xx (xx.x%) |
| | (%x xx) xx |

Denominator of percentage is number of subjects screened.

| Version: 4.0 | Confidential |
|---------------------|--------------|
| Date: Mar 5th, 2023 | |

| Age Men (SD) | Mean (SD) | | Statistics | Group 1<br>(N=) | Group 2 $(N=)$ | Group 3 $(N=)$ | Group 4<br>(N=) | Group 5 $(N=)$ | Overall (N=) |
|---|---|---|---|---|---|---|---|---|---|
| au (SD) dedian 2), Q3 iii, Max iii, Max (xx.x%) | au (SD) dedian 21, Q3 in, Max n (%) (xx.x%) | Ασο | r | | | | | | |
| an (SU) // dedian // dedian // do) // (Xx.X%) | an (SD) // dedian // dedian // (%) // (Xx,x%) // (Xx,x | 200 | 1 | | | | | | |
| 4 c dian 4 c dian 4 c dian 4 c dian 5 l . Q 3 2 l . Q 3 2 l . Q | 4edian 31, Q3 iii, Max iii, Max iii, Max (xx.x%) | | Mean (SD) | | | | | | |
| 21, Q3 iii, Max iii, Max iii, Max (xx.x%) | 21, Q3 iii, Max iii, May iii, Ma, iii, May iii, Max iii, | | Median | | | | | | |
| 11 (%) (Xx, x, x | 11, Max 11 (%) (xx, x%) | | 01 03 | | | | | | |
| II, Max | III, Max II (%) (XX.X%) | | 5,5 | | | | | | |
| 11 (%) (XX.X%) | 11 (%)<br>(xx.x%) | | Mın, Max | | | | | | |
| (''''') ('''''''''''''''''''''''''''''''''''' | 11(%) (XXX%) | | ( e | | | | | | |
| (Xx, x, y, o) | (Xx, x, y, 0)<br>(Xx, x | Sex | n (%) | | | | | | |
| (XXX%) | (XXX%) | Female | xx(xx.x%) | | | | | | |
| (XXX%) | 1 (%)<br>(XX, 2%) | Male | (%x.xx)xx | | | | | | |
| 11(%)<br>(Xx, 2%) | (%α)<br> (%αχ%)<br> (% | | į | | | | | | |
| (Xx, x%)<br>(Xx, x | (Xx, x%)<br>(Xx | Ethnicity | n (%) | | | | | | |
| (XX.X%) | (XX.X%) | Luo | xx(xx.x%) | | | | | | |
| (xx x%) | (XXX%) | Luhya | xx(xx.x%) | | | | | | |
| (xx x%) | (xx x%) | Not reported | (%x.xx)xx | | | | | | |
| n(%)<br>(XXX%) | (XXX%) | Thenoun | (%0 x x)xx | | | | | | |
| (XXX%) | (XXX%) | Olikilowii | (0/Y'YY)YY | | | | | | |
| 11 (%) (XX.X%) | n (%)<br>(xx x%) | Other | xx(xx.x%) | | | | | | |
| (XXX%) | (XXX%) | Race | n (%) | | | | | | |
| (XXXX%) | (XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | White | (%)0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 0 | | | | | | |
| (XXXX%) | (XX,X%) | w IIIC | (0/v:vv)vv | | | | | | |
| (XX.X%) | (XX,X%) | Black | XX(XX.X%) | | | | | | |
| (XXX%) | (Xx, x, y, 0)<br>(Xx, x | Not reported | xx(xx.x%) | | | | | | |
| (Xx, X%) (X, X%) | (XX X%) | Unknown | xx(xx.x%) | | | | | | |
| (xx.x%) | (Xx, x%) | Other | xx(xx.x%) | | | | | | |
| 10(%) (XX.X%) | 10(%) (Xx.x%) | | Š | | | | | | |
| (xx,x%) | (XXX%) | HIV Status | n(%) | | | | | | |
| (Xx, x%) | (XXX%) | Positive | xx(xx.x%) | | | | | | |
| n (%) (xx.x%) | (xx.x%) | Negative | (%X.XX)XX | | | | | | |
| (xx.x%) | (XXX%) | Own Bednet? | n (%) | | | | | | |
| (xx.x%)<br>(xx.x%)<br>(xx.x%)<br>(xx.x%)<br>(xx.x%)<br>(xx.x%)<br>(xx.x%) | (xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%)<br>(xxx%) | Yes | (%x:xx)xx | | | | | | |
| (xx,x%)<br>(xx,x%)<br>(xx,x%)<br>(xx,x%)<br>(xx,x%)<br>(xx,x%) | n (%)<br>(xx,x%)<br>(xx,x%)<br>(xx,x%)<br>(xx,x%)<br>(xx,x%) | No | xx(xx.x%) | | | | | | |
| (XXX%)<br>(XXX%)<br>(XXXX%)<br>(XXXX%)<br>(XXXX%)<br>(XXXX%) | (XXX%)<br>(XXX%)<br>(XXX%)<br>(XXX%)<br>(XXXX%)<br>(XXXX%) | Sleen Under Not? | (%) u | | | | | | |
| (xx.x%) (xx.x%) (xx.x%) (xx.x%) (xx.x%) | (XXX%) (XXX%) (XXX%) (XXX%) (XXX%) (XXX%) | Vee | (0/) = | | | | | | |
| (XXX%) (XXX%) (XXX%) (XXX%) (XXX%) | (XXX%)<br>(XXX%)<br>(XXX%)<br>(XXX%)<br>(XXX%) | 1.03 | (0/ 2/24) | | | | | | |
| (XX,X%) (XX,X%) (XX,X%) | (Xx,x%)<br>(Xx,x%)<br>(Xx,x%) | Опсе а week | XX(XX.X%) | | | | | | |
| (XX,X%) (XX,X%) | (XX,X%) (XX,X%) | 2-3 times a week | xx(xx.x%) | | | | | | |
| (Xx x%) (Xx x%) | (XX,X%) (XX,X%) | 4-6 times a week | xx(xx.x%) | | | | | | |
| (xx.x%) | (xx.x%) | Daily | xx(xx.x%) | | | | | | |
| | | No | XX(XX.X%) | | | | | | |
| | | Persion: 4.0 | | | | | | onfident | ial |
| LALL WALL BALL 11111 | vate: Mar 5th. 2023 | CISIOII. 4.0 | | | | | , | VIIIIACIII | 141 |


| | | | | | | | | | | Indoor residual | n (%) |
|---|---|---|---|---|---|---|---|---|---|---|---|
| xx(xx.x%) xx(xx.x%) n Mean (SD) Median Q1, Q3 | xx(xx.x%) xx(xx.x%) n Mean (SD) Median Q1, Q3 Min, Max | xx(xx.x%) xx(xx.x%) n Mean (SD) Median Q1, Q3 Min, Max n | xx(xx.x%) xx(xx.x%) n Mean (SD) Median Q1, Q3 Min, Max n Mean (SD) | xx(xx.x%) xx(xx.x%) n Mean (SD) Median Q1, Q3 Min, Max n Mean (SD) Median | xx(xx.x%) xx(xx.x%) n Mean (SD) Median Q1, Q3 Min, Max n Mean (SD) Median Q1, Q3 | xx(xx.x%) xx(xx.x%) n Mean (SD) Median Q1, Q3 Min, Max n Median Q1, Q3 Median Q1, Q3 Min, Max | xx(xx.x%) xx(xx.x%) n Mean (SD) Median Q1, Q3 Min, Max n Median Q1, Q3 Min, Max n n n n n n n n n n n n n | xx(xx.x%) xx(xx.x%) n Mean (SD) Median Q1, Q3 Min, Max n Median Q1, Q3 Min, Max n Median Q1, Q3 Min, Max | xx(xx.x%) n Mean (SD) Median Q1, Q3 Min, Max n Mean (SD) Median Q1, Q3 Min, Max n Median Q1, Q3 Min, Max | spray within the past<br>year | |
| | | | | | | | | | | | xx(xx.x%) |
| | | | | | | | | | | No | xx(xx.x%) |
| Mean (SD)<br>Median<br>Q1, Q3 | Mean (SD) Median Q1, Q3 Min, Max | | | | | | | | | Height | п |
| Median<br>Q1, Q3 | Median<br>Q1, Q3<br>Min, Max | | | | | | | | | | Mean (SD) |
| 01,03 | Q1, Q3<br>Min, Max | | | | | | | | | | Median |
| | Min, Max | Min, Max<br>Weight n | | | | | | | | | 01,03 |
| | Mean (SD) Median Q1, Q3 Min, Max | Median Q1, Q3 Min, Max n Mean (SD) Median Q1, Q3 | Q1, Q3 Min, Max n Mean (SD) Median Q1, Q3 | Min, Max<br>n<br>Mean (SD)<br>Median<br>Q1, Q3 | n<br>Mean (SD)<br>Median<br>Q1, Q3 | Mean (SD)<br>Median<br>Q1, Q3 | Median<br>Q1, Q3 | Q1, Q3 | | | Min, Max |

N: total number of subjects in each group
n: total number of subjects in each category
Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials to clear parasites; Group 7: Rabies with anti-malarials to clear parasites.


| Z | |
|---------------|---|
| Ą | |
| S | |
| Z | |
| ANALYSIS PLAN | |
| Z | |
| LICAL | |
| S | |
| STATIST | |
| S | |
| fy: | ١ |

| | Group 1 Group 2 Group 3 Gro<br>(N=) $(N=)$ $(N=)$ $(N=)$ $(N=)$ | Group 2<br>(N=) | Group 3<br>(N=) | Group 4<br>(N=) | Group 4 Group 5 (N=) (N=) | Overall (N=) |
|---|---|---|---|---|---|---|
| HLA subtype 1: xxxx | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| HLA subtype 2: xxxx | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |
| HLA subtype 3: xxxx | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) | xx(xx.x%) |

2 subtypes

N: total number of subjects in each group

Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).


STATISTICAL ANALYSIS PLAN

| Table 10.1.5: Protocol Deviations | | | | | | |
|---|---|---|---|---|---|---|
| Protocol Deviation Type/classification | Group 1<br>(N=) | Group 2<br>(N=) | Group 3<br>(N=) | Group 4<br>(N=) | Group 5<br>(N=) | Total<br>(N=) |
| | (%X.XX) XX | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Antimalarial drugs administered incorrectly | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| P administered incorrectly | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Procedure done incorrectly | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) |

| Major $xx(xx.x\%)$ $xx(xx.x\%)$ $xx(xx.x\%)$ $xx(xx.x\%)$ $xx(xx.x\%)$ $xx(xx.x\%)$ Minor $xx(xx.x\%)$ $xx(xx.x\%)$ $xx(xx.x\%)$ $xx(xx.x\%)$ | Deviation Classifications | | | | | | |
|---|---|---|---|---|---|---|---|
| XX (XX.X%) $XX (XX.X%)$ $XX (XX.X%)$ $XX (XX.X%)$ | Major | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Minor | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |

N: total number of subjects in each group
Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials to clear parasites.


| Table 10.1.6: Medical History | ledical History | | | | | |
|---|---|---|---|---|---|---|
| System Organ Class/ | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total |
| Preferred Term | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) |
| System Organ Class #1 | | | | | | |
| Preferred term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #2 | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx |
| :: | : | : | : | : | : | : |
| System Organ Class #2 | | | | | | |
| Preferred term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| : | : | : | : | : | : | : |
| System Organ Class #3 | | | | | | |
| Preferred term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx |
| | : | : | : | : | : | : |

N: total number of subjects in each group
Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials with anti-malarials with a group for the formula for the formu

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis). N: total number of subjects in each group


| | , | • | • | | | |
|---|---|---|---|---|---|---|
| Body System | Group I<br>(N=) | Group 2<br>(N=) | Group 3<br>(N=) | Group 4<br>(N=) | Group 5<br>(N=) | (N=) |
| General appearance at Visit 5 | | | | | | |
| Normal | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not done | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| General appearance Visit 11 | | | | | | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not done | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| General appearance at Visit 17 | | | | | | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Abnormal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Not done | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) |

(Display additional rows for the other categories of physical

exam)

N: total number of subjects in each group

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

The physical examination includes the following body system or part: 1. General appearance; 2. Skin; 3. Lymph nodes; 4. HEENT; 5. Neck; 6. Respiratory/pulmonary; 7. Cardiovascular; 8. Abdomen; 9. Musculoskeletal; 10. Neurological; 11. Extremities; 12. Other


| Table 10.1.9: Prior Medications | Medications | | | | | |
|---|---|---|---|---|---|---|
| ATC Level/ Preferred Term | Group 1<br>(N=) | Group 2<br>(N=) | Group 3<br>(N=) | Group 4<br>(N=) | Group 5<br>(N=) | Total<br>(N=) |
| ATC Classification #1 | | | | | | |
| Preferred term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC Classification #2 | | | | | | |
| Preferred term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ATC Classification #3 | | | | | | |
| Preferred term #1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Preferred term #3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| : | | | | | | : |

N: total number of subjects in each group
Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials with anti-malarials with a group for the formula for the formu

Document ID: 2940b9f833d20dadf1251001aa420c67b5b7d78213e65c8226c47e70a74c3f5a


| | Total<br>(N=) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Group 5<br>(N=) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Group 4<br>(N=) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | (%XXX) XX | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | Group 3 $(N=)$ | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ations | Group 2 $(N=)$ | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| omitant Medic | Group 1<br>(N=) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Table 10.1.10: Concomitant Medications | ATC Level/ Preferred Term | ATC Classification #1 | Preferred term #1 | Preferred term #2 | Preferred term #3 | ATC Classification #2 | Preferred term #1 | Preferred term #2 | Preferred term #3 | ATC Classification #3 | Preferred term #1 | Preferred term #2 | Preferred term #3 |

N: total number of subjects in each group Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials to clear parasites.


| z |
|-----------------|
| Ā |
| $\sim$ |
| YSIS PLAN |
| _ |
| STATISTICAL ANA |
| ď |
| Ā |
| $\Gamma$ |
| 2 |
| M |
| S |
| ы |

| Table | Table 10.1.11: Vaccine Administration | Administration | | |
|---|---|---|---|---|
| Group | Visit 5-Dosel | Visit 11-Dose2 | Visit 17-Dose3 | # of subjects<br>who received<br>all three<br>vaccine doses |
| Group 1 (N=) xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 2 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 3 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 4 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 5 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Total | (% x x x) xx | (% x xx) xx | (% x xx) xx | (% x xx) xx |

Total xx (xxx. %) xx (xxx. %) xx (xxx. %) xx (xxx. %)

N: total number of subjects in each group

N: total number of subjects in each group

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to pervent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials treatment to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarial to clear parasites; Group 5: Rabies with anti-malarial to clear parasites; Group 5: Rabies


Table 10.1.12: Anti-Malarial Compliance

| | x) xx |
|-------|------------------------------------------|
| × × × | (% ( |
| x (%x | XX (XXX |

xx: represents the number of subjects who took the full dose of anti-malarials.

N: total number of subjects in each group

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 4: Rabies with anti-malarials to clear parasites. Group 5: Rabies with anti-malarials to prevent infection (prophylaxis)

Stables with anti-malarials to prevent infection (prophylaxis)

HA/Pip: Dihydroartemisinin-piperaquine; LD PQ: Low dose primaquine; AL: Artemether/lumefantrine (Coartem)

TABLE 10.1.13.1: VISIT ATTENDANCE (EPOCH 1)

| i | | | | Trea | Freatment and immunoization (Epoch 1) | ınoization (Epoc | ch 1) | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Group | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 | : | Repeat until<br>Visit 18 |
| Group 1 (N=) | Group 1 (N=) xx (xx.x %) | xx (xx.x %) | xx (xx.x %) xx (xx.x %) | xx (xx.x %) | xx (xx.x %) xx (xx.x %) | xx (xx.x %) | xx (xx.x %) xx (xx.x %) | xx (xx.x %) | | |
| Group 2 (N=) | Group 2 (N=) xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | | |
| Group 3 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | | |
| Group 4 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | | |
| Group 5 (N=) | xx (xx.x %) | xx (xx.x %) | (% x.xx) xx | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | | |
| Total | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | | |

N: total number of subjects in each group
Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis); Group 4: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials with anti-malarials with anti-malarials with a transfer with a transfe

 Date: Mar 5th, 2023

TABLE 10.1.13.2: VISIT ATTENDANCE (EPOCH 2)

| Ç | | | | Active Deta | Active Detection of Infection (Epoch 2) | n (Epoch 2) | | | |
|---|---|---|---|---|---|---|---|---|---|
| dronb | Visit 19 | Visit 20 | Visit 21 | Visit 22 | Visit 23 | Visit 24 | Visit 25 | Visit 26 | Visit 27 |
| Group 1 (N=) | xx (xx.x %) | Group 1 (N=) $xx (xx.x \%)$ $xx (xx.x \%)$ | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) xx (xx.x %) xx (xx.x %) | xx (xx.x %) | (% x.xx) xx | xx (xx.x %) | (% x.xx) xx |
| Group 2 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 3 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 4 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 5 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Total | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

N: total number of subjects in each group
Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials with anti-malarials with a group 6: Rabies wit

 Date: Mar 5th, 2023

TABLE 10.1.13.3: VISIT ATTENDANCE (EPOCH 3)

| | | | | Active Detection of Infection-Extension (Epoch 3) | of Infection-Ext | ension (Epoch 3) | ( | |
|---|---|---|---|---|---|---|---|---|
| Group | Visit 28 | Visit 29 | Visit 30 | | Visit 31 Visit 32 | Visit 33 | Visit 34 | Visit 35 |
| Group 1 (N=) | xx (xx.x %) | Group I (N=) $xx (xxx. \%)$ $xx (xxx. \%)$ $xx (xxx. \%)$ $xx (xxx. \%)$ $xx (xxx. \%)$ | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 2 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 3 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |
| Group 4 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | (% x.xx) xx | xx (xx.x %) |
| Group 5 (N=) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | (% x.xx) xx | xx (xx.x %) |
| Total | xx (xx.x %) | xx (xx.x %) xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) | xx (xx.x %) |

N: total number of subjects in each group
Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials with a group for factor of the factor of


#### VACCINE EFFICACY TABLES

Table 10.2.1.1 and 2. Vaccine efficacy (Group 1 vs Group 4): First Infection Events (FIEs) of P. falciparum during the Active Detection of Infection period by HIV status and overall (ATP cohort for efficacy and Total cohort for efficacy)

| First or only infection | | Group 1 | Group 1 (RTS,S) | | Grou | Group 4 (Rabies) | ies) | | | Vaccine | Vaccine Efficacy | | Adjusting<br>variable | Interaction VE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | z | Events | PYAR | Rate | z | Event | PYAR | N Events PYAR Rate N Event PYAR Rate | | TT | UL | P value | Efficacy LL UL P value P value | P value |
| Overall<br>unadjusted | XXX | xxx | XXXX.X X.XX | X.XX | XXX | XXX XXX | XXX | XXXX.X | XX.XX | XX.XX XX.XX | | X.XXX | | |
| Adjusted by HIV | | | | | | | | | XX.XX | XX.XX | xx.xx | X.XXX | X.XXX | X.XXX |
| HIV positive | ×× | XXX | XXXXXX X.X | X.X | ×× | XXX | XXX | XXXX.X | | | | | | |
| HIV negative Xxx xxx | XX | XXX | XXXX.X X.X | X.X | XXX | XXX XXX | XXX | XXXX.X | | | | | | |

N = total number of subjects at risk in each group (without missing values) Events = number of subjects having at least one confirmed P. falciparum infection detected by PCR in each group PYAR = sum of follow-up period (censored at the first occurrence of a confirmed P. falciparum infection) expressed in years

Events/PYAR = Incidence rate of subjects reporting one event LL, UL = 95% Lower and Upper confidence limits

Efficacy (%) = Vaccine Efficacy adjusted by gender (Cox regression model, 1-adjusted HR (Hazard ratio))

For the multivariable analysis, HIV (positive vs negative) will be included, and the next variables will be considered: Age (tertile 1-3), Gender (male vs female), the more significant between Ethnicity p-values for vaccine efficacy and statistically significant covariates are from Cox regression model and interaction vaccine efficacy p-value is from HIV status and treatment Group term.

and Race, the most significant between Own bednet, Sleep under bednet and Indoor residual spray (IRS) and the most significant between Height, Weight and BMI (tertile 1-3). Any potential confounding factor will be identified with p-value lower than 0.1.  Date: Mar 5th, 2023

Table 10.2.2.1 and 2 Vaccine efficacy (Group 2 vs Group 5): First Infection Events (FIEs) of P. falciparum during the Active Detection of Infection period by HIV status and overall (ATP cohort for efficacy and Total cohort for efficacy)

| First or only<br>infection | | Group 2 (RTS,S) | (RTS,S) | | Grou | Group 5 (Rabies) | ies) | | | Vaccin | Vaccine Efficacy | | Adjusting<br>variable | Interaction VE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| - | Z | Events | PYAR | N Events PYAR Rate | Z | Event | PYAR | N Event PYAR Rate | Efficacy | TT | nr | P value | Efficacy LL UL P value P value | P value |
| Overall X<br>unadjusted | ×× | Xxx xxx | XXXX.X X.XX | X.XX | xxx xxx | XXX | XXX | XXXX.X | XX.XX | XX.XX | XX.XX XX.XX | X.XXX | | |
| Adjusted by HIV | | | | | | | | | XX.XX | XX.XX | XX.XX | X.XXX | X.XXX | X.XXX |
| HIV positive X | ×× | XXX | XXXXX.X | X.X | XX | XXX | XXX | XXXX.X | | | | | | |
| HIV negative X | ×× | Xxx xxx | XXXXX.X X.X | X.X | XXX XXX | xxx | XXX | XXXX.X | | | | | | |

N = total number of subjects at risk in each group (without missing values)

Events = number of subjects having at least one confirmed P. falciparum infection detected by PCR in each group

PYAR = sum of follow-up period (censored at the first occurrence of a confirmed P. falciparum infection) expressed in years

Events/PYAR = Incidence rate of subjects reporting one event

LL, UL = 95% Lower and Upper confidence limits

Efficacy (%) = Vaccine Efficacy adjusted by gender (Cox regression model, 1-adjusted HR (Hazard ratio))

p-values for vaccine efficacy and statistically significant covariates are from Cox regression model and interaction vaccine efficacy p-value is from HIV status and treatment Group term. For the multivariable analysis, HIV (positive vs negative) will be included, and the next variables will be considered: Age (tertile 1-3), Gender (male vs female), the more significant between Own bednet, Sleep under bednet and Indoor residual spray (IRS) and the most significant between Height, Weight and BMI (tertile 1-3). Any potential

confounding factor will be identified with p-value lower than 0.1.

 Date: Mar 5th, 2023

Table 10.2.3.1 and 2 Vaccine efficacy (Group 1 vs Group 2): First Infection Events (FIEs) of P. falciparum during the Active Detection of Infection period by HIV status and overall (ATP cohort for efficacy and Total cohort for efficacy)

| First or only | | | (S SLAW) | | | one, | 6 | | | Vaccing | Vaccine Efficacy | | Adjusting | Interaction VE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| infection | Z | Group Events | Group I (KI 5,5) Events PYAR | Rate | Z | Group 2 (K.1.3,5) N Event P | PYAR | Group 1 (RUS,5) Group 2 (RUS,5) N Events PYAR Rate N Event PYAR Rate | Efficacy | rr | nr nr | P value | Efficacy LL UL P value P value P value | P value |
| Overall unadjusted | ×× | XXX | XXXX.X | Xxx xxx x.xx x.xx | ×× | XXX XXX | XXX | XXXX.X | XX.XX XX.XX XX.XX | XX.XX | XX.XX | X.XXX | | |
| Adjusted by HIV | | | | | | | | | XX.XX | XX.XX | XX.XX | XXXX | X.XX | X.XXX |
| HIV positive | ×× | XXX | XXXXX.X | X.X | XX | XXX | XXX | XXXX.X | | | | | | |
| HIV negative Xxx | ×× | XXX | XXXX.X X.X | X.X | XX | XXX | XXX | XXXX.X | | | | | | |

N = total number of subjects at risk in each group (without missing values)

Events = number of subjects having at least one confirmed *P. falciparum* infection detected by PCR in each group

PYAR = sum of follow-up period (censored at the first occurrence of a confirmed *P. falciparum* infection) expressed in years

Events/PYAR = Incidence rate of subjects reporting one event

LL, UL = 95% Lower and Upper confidence limits

Efficacy (%) = Vaccine Efficacy adjusted by gender (Cox regression model, 1-adjusted HR (Hazard ratio))

p-value from Cox regression model

For the multivariable analysis, HIV (positive vs negative) will be included, and the next variables will be considered: Age (tertile 1-3), Gender (male vs female), the more significant between Own bednet, Sleep under bednet and Indoor residual spray (IRS) and the most significant between Height, Weight and BMI (tertile 1-3). Any potential confounding factor will be identified with p-value lower than 0.1.

 Date: Mar 5th, 2023

## Protocol No. CVIA-078; RTS,S/AS01 E

STATISTICAL ANALYSIS PLAN

Table 10.2.4.1 and 2 Vaccine efficacy (Group 4 vs Group 5): First Infection Events (FIEs) of P. falciparum during the Active Detection of Infection period by HIV status and overall (ATP cohort for efficacy and Total cohort for efficacy)

| First or only infection | | Group 4 | Group 4 (Rabies) | | Grou | Group 5 (Rabies) | ies) | | | Vaccine | Vaccine Efficacy | | Adjusting<br>variable | Interaction VE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Z | Events | PYAR | Rate | z | Event | PYAR | N Events PYAR Rate N Event PYAR Rate | Efficacy | TT | UL | P value | Efficacy LL UL P value P value P value | P value |
| Overall<br>unadjusted | XX | xxx | XXXX.X | X.XX | XX | xxx | xxx | XXXX.X | XXX XXX XXXXX XXXXX XXXXX XXXXX XXXXX XXXX | XX.XX | XX.XX | X.XXX | | |
| Adjusted by HIV | | | | | | | | | XX.XX | XX.XX | XX.XX XX.XX | X.X.X | X.XX.X | X.XXX |
| HIV positive | ×× | XXX XXX | XXXXXX X.X | X.X | XXX XXX | XXX | XXX | XXXX.X | | | | | | |
| HIV negative Xxx xxx | ×× | xxx | XXXX.X | xxx x.x | XX | xxx xxx | XXX | XXXX.X | | | | | | |

N = total number of subjects at risk in each group (without missing values)

PYAR = sum of follow-up period (censored at the first occurrence of a confirmed P. falciparum infection) expressed in years Events = number of subjects having at least one confirmed P. falciparum infection detected by PCR in each group

Events/PYAR = Incidence rate of subjects reporting one event

LL, UL = 95% Lower and Upper confidence limits

Efficacy (%) = Vaccine Efficacy adjusted by gender (Cox regression model, 1-adjusted HR (Hazard ratio))

p-value from Cox regression model

For the multivariable analysis, HIV (positive vs negative) will be included, and the next variables will be considered: Age (tertile 1-3), Gender (male vs female), the more significant between Own bednet, Sleep under bednet and Indoor residual spray (IRS) and the most significant between Height, Weight and BMI (tertile 1-3). Any potential confounding factor will be identified with p-value lower than 0.1.


# Protocol No. CVIA-078; RTS,S/AS01<sub>E</sub> STATISTICAL ANALYSIS PLAN

Table 10.2.5.1 and 2 Summary of subjects at risk, person-time, number of FIEs and incidence rate (ATP cohort for efficacy and Total cohort for efficacy) for Group 1 and 4

| | | Group 1 | Group 1 (RTS/S) | | | Group 4 | Group 4 (Rabies) | | | 000 | Overall | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Z | Events | PYAR | Rate | Z | Events | PYAR | Rate | Z | Events | PYAR | Rate |
| Visit 19 | Xxx | XX | XX.X | X.X | XXX | XX | XX.X | X.X | XXX | xx | XX.X | X.X |
| Visit 20 | Xxx | XX | xx.x | X.X | XXX | xx | XX.X | X.X | XXX | XX | XX.X | X.X |
| Visit 21 | Xxx | XX | XX.X | X.X | XXX | XX | XX.X | X.X | XXX | XX | XX.X | X.X |
| Visit 22 | Xxx | XX | xx.x | X.X | XXX | xx | XX.X | X.X | XXX | XX | XX.X | x.x |
| Visit 23 | Xxx | XX | XX.X | X.X | XXX | XX | XX.X | X.X | XXX | XX | XX.X | X.X |
| Visit 24 | XXX | X | XX.X | X.X | XXX | XX | XX.X | X.X | XXX | XX | XX.X | x.x |
| Visit 25 | XXX | XX | XX.X | X.X | XXX | XX | XX.X | X.X | XXX | XX | XX.X | x.x |
| Visit 26 | XXX | XX | XX.X | X.X | XXX | XX | XX.X | X.X | XXX | XX | XX.X | X.X |
| Visit 27 | XXX | XX | XX.X | X.X | XXX | XX | XX.X | X.X | XXX | XX | XX.X | X.X |
| Fig. 1. The targets are not reach by the end of Epoch 2, then ADI period will extended to when the target is reached or the end of the extension ADI period NII period NII extension ADI period NII period will extension ADI period NIII | at risk in ee | ach group at ea | ıch visit (with | guissing moon | values) | | | | | | | |
| Events = number of subjects having at least one confirmed <i>P. falciparum</i> infection detected by PCR PCR PVAR = sum of follow-up period (censored at the first occurrence of a confirmed <i>P. falciparum</i> infection) expressed in years | bjects havm; | g at least one c<br>(censored at the | confirmed P., e first occurre | falciparum 1<br>ince of a cor | nfection deta<br>rfirmed P. fa | ected by PCR<br>dciparum infec | ction) express | sed in years | | | | |
| E | J + | State of the state | *************************************** | _ | | | | | | | | |

Commented [JA1]: Why is this footnote removed?

Events/PYAR = Incidence rate of subjects reporting one event No parasitemia testing has been recorded for unscheduled visits.

Commented [JJ2R1]: There were no parasitemia data for unscheduled visits during ADI

**Commented [JA3R1]:** Could you please include in the footnote that no parasitemia data for unscheduled visits was registered.

Please note that there are several AEs that are malaria, but I have not check if they were during the ADI epochs.

Commented [JJ4R1]: Updated


| 15 |
|--------|
| 2 and |
| roup |
| or G |
| cy) f |
| effica |
| for |
| hort |
| tal co |
| d To |
| y an |
| fficac |
| or ef |
| ort f |
| P coh |
| (ATF |
| rate |
| ence |
| incid |
| and |
| FIES |
| r of |
| umbe |
| ne, n |
| n-tir |
| perso |
| risk, |
| ts at |
| ubjec |
| of su |
| mary |
| Sum |
| nd 2 |
| 6.1 an |
| 10.7 |
| able |
| Ξ |

| | | Group 2 | Group 2 (RTS/S) | | | Group 5 | Group 5 (Rabies) | | | )<br>O | Overall | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Z | Events | PYAR | Rate | Z | Events | PYAR | Rate | Z | Events | PYAR | Rate |
| Visit 19 | XXX | | | | XXX | | | | XXX | | | |
| Visit 20 | XXX | XX | XX.X | X.X | XXX | xx | XX.X | X.X | XXX | XX | XX.X | x.x |
| Visit 21 | XXX | XX | XX.X | X.X | XXX | xx | XX.X | X.X | XXX | XX | XX.X | x.x |
| Visit 22 | XXX | XX | XX.X | X.X | XXX | xx | XX.X | X.X | XXX | XX | XX.X | x.x |
| Visit 23 | XXX | XX | XX.X | X.X | XXX | xx | XX.X | X.X | XXX | XX | XX.X | x.x |
| Visit 24 | XXX | XX | XX.X | X.X | XXX | xx | XX.X | X.X | XXX | XX | XX.X | X.X |
| Visit 25 | XXX | xx | XX.X | X.X | XXX | xx | XX.X | X.X | XXX | XX | XX.X | x.x |
| Visit 26 | XXX | XX | XX.X | X.X | XXX | xx | XX.X | X.X | XXX | XX | XX.X | x.x |
| Visit 27 | xxx | X | xx.x | X.X | xxx | xx | x.x.x | x.x | xxx | X | x.x.x | X.X |
| : | | | | | | | | | | | | |
| If the targets are not | | | | | | | | | | | | |
| reach by the end of | | | | | | | | | | | | |
| Epoch 2, then ADI | | | | | | | | | | | | |
| period will | | | | | | | | | | | | |
| extended to when | | | | | | | | | | | | |
| the target is reached | | | | | | | | | | | | |
| or the end of the | | | | | | | | | | | | |
| extension ADI | | | | | | | | | | | | |

N = number of subjects at risk in each group at each visit (without missing values)

Events = number of subjects having at least one confirmed *P. falciparum* infection detected by PCR

PYAR = sum of follow-up period (censored at the first occurrence of a confirmed *P. falciparum* infection) expressed in years

Events/PYAR = Incidence rate of subjects reporting one event

No parasitemia testing has been recorded for unscheduled visits.

period


# Protocol No. CVIA-078; RTS,S/AS01 E STATISTICAL ANALYSIS PLAN

Table 10.2.7.1 and 2 Summary of median time to FIEs and hazards (ATP cohort for efficacy and Total cohort for efficacy)

| | Group1 (IN=) | Croup2 (IN=) | Group4 (N=) | Croups (N=) | Overall (N=) |
|---|---|---|---|---|---|
| Median time to FIEs (IQR) | XXX(XXX.X-XXX.X) | xxx(xxx.x-xxx.x) | xxx(xxx.x-xxx.x) | (X.XXX.X.XXXXXX) | XXX(XXX.X-XXX.X) |
| Hazard (95% CI) | X.XX(X.XX-X.XX) | X.XX(X.XX-XXXX) | X.XX(X.XX-X.XX) | X.XX(X.XX-X.XX) | X.XX(X.XX-XXX) |

N=number of subjects at risk in each group (without missing values) Median time to FIEs (expressed in years) and hazard are derived from KM and cox regression model respectively.


#### IMMUNOGENICITY TABLES

MTs (ATP cohort for immunogenicity

| | | | Group 1 | Group 2 | Group 3 |
|---|---|---|---|---|---|
| Anti-CS NANP<br>(1XPBS) | Visit | Statistics | | | |
| sei oi esponse | Visit 2 | z | XX | × | XX |
| | | z | XX | XX | Xx |
| | | % | XX.X | x.xx | XX.X |
| | | LL, UL | XX.X | XX.X | XX.X |
| | Repeat for visits 11, 13, 17, 10 and 27 and the termination visit | | | | |
| Repeat for<br>Anti-CS NANP<br>(4M Urea) | | | | | |
| Anti-CS NANP<br>(1XPBS) GMT | | | | | |
| | Visit 2 | Titer | xxx.x | XXX.X | XXX.X |
| | | LL, UL | XXX-XX-XXX | XXX.XX- | XXX.XX-<br>XX.X |
| | | Min, Max | XXXX-XXXXX | XXXX.X- | XXX.X- |
| | | p-value | 1 vs 2 | 2 vs 3 | 1 vs 3 |
| | Repeat for visits 11, 13, 17, 10 and 27 and the termination visit | | (vvv·v) | (vvv <sup>(</sup> v) | (vvv:v) |
| Repeat for<br>Anti-CS NANP<br>(4M Urea)<br>GMT and | | | | | |


#### Anti-CS NANP Avidity Index

Abbreviations: GMT = Geometric Mean Titor; N = Total number of subjects; n = Number of seropositive subjects; % = Percentage; LL = Lower limit of 95% CI; UL = Upper limit of 95% CI; Min = Minimum; Max = Maximum;

p-values for pairwise comparisons are computed from mixed model for repeated measures using avidity index or log transformed antibody titers (Anti-CS NANP (1XPBS) and Anti-CS NANP (4M Urea)) and their interaction term as dependent variables and groups and HIV status as covariates and subject as random effect.

Seropositivity criteria: antibody titer > LLOQ, lower limit of quantification

Table 10,3.2.1 and 2: Number and Percentage of Subjects with Anti-CS C-term Antibody Titer/Avidity Equal to or above Cut-off and GMTs (ATP cohort for immunogenicity and Same shell as T.10.3.1

Table 10.3.3.1 and 2: Number and Percentage of Subjects with Anti-H8sAb Titer Equal to or above Cut-off and GMTs (ATP cohort for immunogenicity and Total vaccinated

Same shell as T.10.3.1 except only antibody titer is assayed and the visits are 2, 5, 11 and 20.


Date: Mar 5th, 2023

# Protocol No. CVIA-078; RTS,S/AS01 E STATISTICAL ANALYSIS PLAN

Table 10.3.4.1 and 2: Geometric Fold Rise in Anti-CS NANP Antibody Titer at Each Post-Vaccination Timepoint Compared to Screening (ATP cohort for immunogenicity and Total vaccinated cohort)

| ntibody Group | | | | | | | 95% CI | D, | | >= 2 | | | >= 3 | | | >= <del>4</del> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | z | Visit | GMT | T Baseline<br>GMT | Ratio<br>Order | Ratio<br>Value | TT | LL UL n | п | %<br>(95% CI) | p-<br>value | п | %<br>(95% CI) | p-<br>value | п | % p- n- % (95% CI) p-value (95% CI) | p-value |
| Anti-CS<br>NANP | | V111 | XX.X | XX.X | V11/V5 | xx.x | XX.X | xxx xx | XX | XX.X (XX.X, XX.X) | 1 vs 2<br>(x.xxx) | × | _ | 1 vs 2<br>(x.xxx) | × | 1 vs 2<br>xx.x(xx.x, xx.x) (x.xxx) | 1 vs 2<br>(x.xxx) |
| 2 | | V111 | XX.X | XX.X | V11/V5 | XX.X | XXX XXXX | XX.X | × | xx.x<br>(xx.x, xx.x) | 2 vs 3 (x.xxx) | X | XX.X<br>(XX.X, XX.X) | 2 vs 3 (x.xxx) | xx | XX.X(XX.X, XX.X) | 2 vs 3<br>(x.xxx) |
| т | | V11 | XX.X | XX.X | V11/V5 | XX.X | XX.X | XX.X | × | xx.x<br>(xx.x, xx.x) | 1 vs 3<br>(x.xxx) | × | (xx.x, xx.x) (x | 1 vs 3<br>(x.xxx) | XX | xx.x(xx.x, xx.x) | 1 vs 3<br>(x.xxx) |
| Repeat for visits 13, | | | | | | | | | | | | | | | | | |
| 17, 10 and 27 and the termination | | | | | | | | | | | | | | | | | |

Abbreviations: GMT = Geometric Mean Titer; N = Total number of subjects; n = Number of seropositive subjects; % = Percentage; LL = Lower limit of 95% CI; UL = Upper limit of 95% CI; Min = Minimum; Max = Maximum;

p-values for pairwise comparisons are computed from mixed model for repeated measures using log transformed fold increase (Anti-CS NANP (1XPBS) and Anti-CS NANP (4M Urea)) and their interaction term as dependent variables and groups and HIV status as covariates and subject as random effect; >=2, >=3 and >=4 responder rates and their 95% CIs are calculated through Clopper-Pearson method and p-values are calculated through Fisher's test or Chi-Square test.

Table 10.3.5.1 and 2: Geometric Fold Rise in Anti-CS C-term Antibody Titer at Each Post-Vaccination Timepoint Compared to Screening (ATP cohort for immunogenicity and Total vaccinated cohort)

Same shell as T.10.3.4.1 and 2

Table 10.3.6.1 and 2: Geometric Fold Rise in Anti-HBsAb Titer at Each Post-Vaccination Timepoint Compared to Screening (ATP cohort for immunogenicity and Total vaccinated cohort)
Same shell as T.10.3.4.1 and 2  Date: Mar 5th, 2023 Version: 4.0

#### SAFETY TABLES

Table 10.4.1.1: Overall Safety Profile by Treatment (Safety Population)

| | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total |
|---|---|---|---|---|---|---|
| | (N=) | (N=) | (N=) | (N=) | (N = 1) | (N=) |
| | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] |
| Number of Local Solicited Adverse Events | XXX | XXX | xxx | xxx | xxx | XXX |
| Number of Subjects with any Local Solicited | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Events | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Number of Systemic Solicited Adverse Events | XXX | XXX | XXX | XXX | XXX | XXX |
| Number of Subjects with any Systemic | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Solicited Adverse Events | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Number of Unsolicited Adverse Events | XXX | XXX | XXX | XXX | XXX | XXX |
| Number of Subjects with any Unsolicited | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Adverse Events | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Number of Adverse Events of Special Interest (AFSIs) | XXX | XXX | XXX | XXX | XXX | XXX |
| Number of Subjects with any Adverse Events | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| of Special Interest (AESIs) | [xx.x-xxx] | [xx.x-xxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxx] |
| Number of Serious Adverse Events (SAEs) | XXX | XXX | XXX | xxx | xxx | XXX |
| Number of Subjects with any Serious Adverse | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Events (SAEs) | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxx] | [x.x.x.x.x] [x.x.x.x.x] [x.x.x.x.x] | [xxx-xxx] | [xxx-xxx] |

N: total number of subjects in each group; n = Number of subjects; %= Percentage; C1 = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

All confidence intervals are two-sided 95% via Clopper-Pearson method.

Denominator for percentage is subjects in safety population.


## Protocol No. CVIA-078; RTS,S/AS01 $_{\rm E}$

STATISTICAL ANALYSIS PLAN

Table 10.4.1.2: Frequency of Local Solicited Adverse Events by Treatment and Severity (Safety Population)

| (N=) | | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total |
|---|---|---|---|---|---|---|---|
| N(%) CI | | (N=) | (N=1) | (N=) | (N=) | (N=) | (N=) |
| (%,x,x,x) | | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] |
| | Any Events | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX(XXX%) XX(XXXX%) XX(XXX%) XX(XXX%) XX(XXX%) XX(XXXX%) XX(XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | [xx.x-xxx] | [xxx-xxx] | [xxx-xxx] | [xx.x-xxx] | [xx.x-xxx] | [xx.x-xxx] |
| XXX-XXX XXX- | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX (XXX%) XX (XXXX%) XX (XXXXX%) XX (XXXXX%) XX (XXXXX%) XX (XXXXX%) XX (XXXXX%) XX (XXXXXX) XX (XXXXXX) XX (XXXXX%) XX (XXXXXX) XX (XXXXXX) XX (XXXXXX) XX (XXXXXXX) XX (XXXXXXX) XX (XXXXXXXX | | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] | [xx.x-xx.x] |
| XX.~XX.4 XXX.~XX.4 XXX.~XX.4 XXX.~XX.4 XXX.XX.6 X | Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX (XXX%) XX (XXXX%) XX (XXXX%) XX (XXXX%) XX (XXXX%) XX (XXXX%) XX (XXXX%) XX (XXXXX) XX (XXXXX) XX (XXXXX) XX (XXXXX) XX (XXXXX) XX (XXXXXX) XX (XXXXXX) XX (XXXXXX) XX (XXXXXX) XX (XXXXXXX) XX (XXXXXXX) XX (XXXXXXXX | | [xx.x-xx.x] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxxx] | [xx.x-xxx] |
| XX.~XX.X XX.~XX.X XX.~XX.X XX.~XX.X XX.XX.86 XX.XX.26 | Grade 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX (XX, X%) XX (XX, X%) XX (XX, X%) XX (XX, X%) | | [xx.x-xx.x] | [xxx-xxxx] | [xxx-xxx] | [xx.x-xxx] | [xx.x-xxx] | [xx.x-xxx] |
| XXXXX XX | Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX (XX X%) XX (XX XX | | [xxx-xxx] | [XXX-XXX] | [xxx-xxxx] | [xxx-xxx] | [xx.x-xx.x] | [xxx-xxx] |
| XX (XX,Y%) | | | | | | | |
| (XX.~XX.X (XX.~XX.X (XX.~XX.X (XX.~XX.X XX (XX.X%) | Pain at SOI | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX (XX X%) | | [xx.x-xxx] | [xxx-xxxx] | [xxx-xxx] | [xx.x-xxx] | [xx.x-xxx] | [xxx-xxx] |
| [XX.*-XX.X] [XX.*-XX.X] [XX.*-XX.X] [XX.*-XX.X] XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) [XX.*-XX.X] [XX.*-XX.X] [XX.*-XX.X] [XX.*-XX.X] XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) XX (XX.X%) [XX.*-XX.X] [XX.*-XX.X] [XX.*-XX.X] [XX.*-XX.X] [XX.*-XX.X] | Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX (XX X%) | | [xx.x-xx.x] | [xxx-xxxx] | [xxx-xxx] | [xx.x-xxx] | [xx.x-xxx] | [xx.x-xxx] |
| [XX.*XX.3] [XX.*XX.3] [XX.*XX.3] [XX.*XX.3] XX(XX.X%) XX(XX.X%) XX(XX.X%) XX(XX.X%) [XX.*XX.3] [XX.*XX.3] [XX.*XX.3] [XX.*XX.3] XX(XX.X%) XX(XX.X%) XX(XX.X%) XX(XX.X%) [XX.*XX.3] [XX.*XX.3] [XX.*XX.3] | Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| XX (XXXX) XX (XXXX) XX (XXXXX) XX (XXXXXX (XXXXX) [XXX-XXX] [XXX-XXX] [XXX-XXX] (XXXXX) XX (XXXXX (XXXXX) (XXX-XXX] (XXX-XXX] [XXX-XXX] [XXX-XXX] | | [xx.x-xxx] | [xxx-xxx] | [xxx-xxx] | [xx.x-xxx] | [xx.x-xxx] | [xx.x-xxx] |
| [XX-XX] [XX-XX] [XX-XX] [XX-XX] XX (XXX/%) XX (XXX/%) XX (XXX/%) XX (XXX/%) XX (XXX/%) [XX-XXX] [XX-XXX] [XX-XXX] | Grade 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| (9%xxx)xx (9%xxx)xx (9%xxx)xx (9%xxx)xx (9%xxx)xx | | [xx.x-xxx] | [xxx-xxx] | [xx.x-xxx] | [xx.x-xx.x] | [xx.x-xxx] | [xx.x-xxx] |
| $[x.xx.x.] \qquad [x.xx.x] \qquad [x.xx.x]$ | Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | | [xx.x-xxx] | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] |

Swelling at SOI)

N: total number of subjects in each group; n = Number of subjects; % = Percentage; CI = Confidence interval.

Group 1: RTS,S/ASOIE with anti-malarials to clear parasites; Group 2: RTS,S/ASOIE with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/ASOIE without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

Denominator for percentage is subjects in safety population.
Subject counted once at highest severity grants.
All confidence intervals are two-sided 95% via Clopper-Pearson method

Local solicited Adverse Events include: Pain at site of injection (Pain at SOI); Swelling at injection site; Each event has intensity scores 0-3 with 0 for no adverse event and 3 for the adverse event that prevents normal activity (for details see protocol for detail)

Date: Mar 5th, 2023


## Protocol No. CVIA-078; RTS,S/AS01E

STATISTICAL ANALYSIS PLAN

Table 10.4.1.3: Frequency of Systemic Solicited Adverse Events by Treatment and Severity (Safety Population)

| | dnomb | 2 dno. | Group 3 | Group 4 | Group 5 | I otal |
|---|---|---|---|---|---|---|
| | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] |
| Any Events | | | | | | |
| Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [x.xx.xx] | [xxx-xxx] | [x.xx.xx] | [x.xx.x] | [xx.x-xx.x] |
| Grade 1 | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] | [xx.x-xxx] |
| Grade 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [xxx-xxx] | [xx.x-xx.x] | [xx.x-xxx] | [xx.x-xxx] | [xx.x-xxx] |
| Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [xx.x-xxx] | [xx.x-xx.x] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] |
| Fever | | | | | | |
| Total | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [x:xx-x:xx] | [x:x-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxx] |
| Grade 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [x.xx.xx] | [xxx-xxx] | [x.xx.xx] | [x.xx.x] | [xx.x-xx.x] |
| Grade 2 | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xx.x-xx.x] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxx] |
| Grade 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | [x.x.x-x.x] | [xxx-xxx] |

(Repeat for Fatigue, Headache, Muscle

ache, and

Gastrointestinal

Symptoms)

N: total number of subjects in each group; n = Number of subjects; % = Percentage; CI = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

Denominator for percentage is subjects in safety population for whom memory aid data was available.

Subject counted once at highest severity grade.

All confidence intervals are two-sided 95% via Clopper-Pearson method

Systemic Solicited Adverse Events include: Fever; Headache; Gastrointestinal symptoms (nausea, vomiting, diarrhea and/or abdominal pain); Fatigue; Muscle ache. Each event has intensity scores 0-3 with 0 for no adverse event and 3 for the adverse event that prevents normal activity. For fever, 0: <37.5°C (99.5°F); 1: 37.5°C (99.5°F) to 38.0°C (100.4°F); 2: >38.0°C (>100.4°F); 0: >38.0°C ( >39.0°C (102.1°F) (for additional details see protocol)


| |
|----------------------------------|

STATISTICAL ANALYSIS PLAN

Protocol No. CVIA-078; RTS,S/AS01  $_{\rm E}$ 

Table 10.4.1.4: Summary of Unsolicited Adverse Events by Treatment (Safety Population)

| | Group 1 $(N=)$ | Group 2 $(N=)$ | Group 3 $(N=)$ | Group 4<br>(N=) | Group 5<br>(N=) | Total<br>(N=) |
|---|---|---|---|---|---|---|
| | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] |
| All Systems | | | | | | |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xx.x-xxx] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| System Organ Class | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 | [xx.x-xxx] | [x.xx.xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [x.x-x.xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xx.x-xxx] | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxx] | [x.xx.xx] | [xxx-xxx] |
| Preferred Term 3 | | | | | | |
| System Organ Class | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | [xxx-xxxx] | [x.x-x.xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [x.x-x.xx] |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [x.xx-x.xx] |
| Preferred Term 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [x:xx-x:xx] | [x.xx-x.xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |

N: total number of subjects in each group; n = Number of subjects; % = Percentage; CI = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

xx= Number of Events Subject counted once per adverse event term. All confidence intervals are two-sided 95% via Clopper-Pearson method.


STATISTICAL ANALYSIS PLAN

Table 10.4.1.5: Summary of Unsolicited Adverse Events by Treatment, Severity and Relationship to Study Treatment (Safety Population)

| | Group 1 | Group 2 | Group 3 | Group 4 | e dno 15 | 10131 |
|---|---|---|---|---|---|---|
| | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] |
| All Systems | | | | | | |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Iotal | [xxx-xxxx] | [x.x.x-x.xx] | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxxx] |
| 1-1-10 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Grade 1 | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] |
| C. C. C. | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Grade 2 | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxxx] |
| C L | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Orade 3 | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] |
| Dolotod | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Kelaled | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxx] | [x:xx-x:xx] | [xx.x-xx.x] |
| 1 4 4 7 | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Olade 1 | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxx] |
| C. F | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Orage 2 | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxx] |
| 2 0000 | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Orade 3 | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxxx] |
| Mot Deleted | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| vot netateu | [xxx-xxx] | [xxx-xxxx] | [xxx-xxxx] | [x.x.x-x.xx] | [xxx-xxxx] | [xxx-xxx] |
| - change | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Olauc 1 | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxxx] |
| Gmda 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Olaue 2 | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxx] |
| Grada 2 | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Orane 3 | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxxx] |
| | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxxx] |
| Carotona Omono Close 1 | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ystem Organ Class 1 | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | [xx.x-xx.x] |
| 10+0 | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| ıotai | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxxx] |
| Carolio 1 | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Orage 1 | [xxx-xxx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [x:xx-x:xx] | [xxx-xxxx] |
| C - | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Grade 2 | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] |


| ) xx (xx.x%) xx (xx.x%) | [ xx.x-xx.x] [xx.x-xx.x] |
|-------------------------|--------------------------|
| xx (xx.x%) | [xxx-xxx] |
| xx (xx.x%) | [xxx-xxx] |
| xx (xx.x%) | [xxx-xxx] |
| (%x.xx) x | [xxx-xxx] |
| XX | |

N: total number of subjects in each group; n = Number of subjects; % = Percentage; CI = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

Xx= Number of Events

All confidence intervals are two-sided 95% via Clopper-Pearson method.

Subjects who experience one or more episodes of the same adverse event are counted once at highest severity grade and relatedness


Table 10.4.1.6: Summary of Serious Adverse Events by Treatment (Safety Population)

| | Group 1<br>(N=) | Group 2 $(N=)$ | Group 3<br>(N=) | Group 4<br>(N=) | Group 5<br>(N=) | Total<br>(N=) |
|---|---|---|---|---|---|---|
| | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] |
| All Systems | | | | | | |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [xxx-xxxx] | [XX.X-XXX.X] | [XX.X-XXX.X] | [XX.X-XXX] | [xxx-xxx] |
| System Organ Class | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 1 | [xx.x-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxxx] |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xx.x-xxx] |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [x.x-x.xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Preferred Term 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [x:xx-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [x:x-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| System Organ Class | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| 2 | [xxx-xxxx] | [x:xx-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [x.xx-x.xx] |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [x.xx.xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [x:x-x:xx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Preferred Term 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |

other SOCs and PTs) (Repeat similarly for

N: total number of subjects in each group; n = Number of subjects; % = Percentage; CI = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabics with anti-malarials to prevent infection (prophylaxis).

XX= Number of Events

Subjects who experience one or more episodes of the same adverse event are counted once
All confidence intervals are two-sided 95% via Clopper-Pearson method.


Table 10.4.1.7: Frequency of Local Solicited Adverse Events by Treatment, Injection Period, and Severity (Safety Population)

| | | Group 1 | | Repeat for Groups 2-5 and |
|---|---|---|---|---|
| | | (N=) | | Total |
| | Injection 1 | Injection 2 | Injection 3 | |
| | Day 1-7 | Day 29-35 | Day 197-203 | |
| | n (%) [CI] | n (%) [CI] | n (%) [CI] | |
| Any Events | (%X.XX) XXX | xxx (xx.x%) | xxx (xx.x%) | |
| | [XX.X-XX.X] | [xx.x-xxx] | [xxx-xxxx] | |
| Total | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [XX.X-XX.X] | [xx.x-xxx] | [xxx-xxxx] | |
| Grade 1 | xxx (xx.x%) | (%x.xx) xxx | xxx (xx.x%) | |
| | [XX.X-XX.X] | [xx.x-xxx] | [xxx-xxxx] | |
| Grade 2 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [XXX-XXXX] | [xx.x-xxx] | [xxx-xxx] | |
| Grade 3 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | |
| Pain at SOI | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxxx] | [xxx-xxxx] | [x.xx-x.xx] | |
| Total | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [XX.X-XX.X] | [xx.x-xxx] | [xxx-xxxx] | |
| Grade 1 | xxx (xx.x%) | (%x.xx) xxx | xxx (xx.x%) | |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] | |
| Grade 2 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [XXX-XXXX] | [xx.x-xxx] | [xxx-xxx] | |
| Grade 3 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxx] | [xxx-xxx] | [x.x.x-xx.x] | |
| Reneat for Swelling at SOD | | | | |

(Repeat for Swelling at SOI)

N: total number of subjects in each group; n = Number of subjects; %= Percentage; CI = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 7: Rabies with anti-malarials to clear parasites; Group 7: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials to clear parasites; Group 7: Rabies with anti-malarial to clear parasites; Group 7: Rabies with anti-malarial to clear parasites; Group 7: Rabies with anti-malarial to clear parasites; Gr

Solicited AEs are collected on the day of vaccine administration and for six days following each injection (Day 1-7). Denominator for percentage is subjects in safety population.

All confidence intervals are two-sided 95% via Clopper-Pearson method.

Local solicited Adverse Events include: Pain at site of injection (Pain at SOI); Swelling at injection site.


| | | Group 1 | | Repeat for |
|------------|-------------|-------------|-----------------|------------|
| | | (N=) | | Groups 2-5 |
| | | | | and Total |
| | Injection 1 | Injection 2 | Injection 3 | |
| | Day 1-7 | Day 29-35 | Day 197-203 | |
| | n (%) [CI] | n (%) [CI] | n (%) [CI] | |
| Any Events | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | |
| Total | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xx.x-xx.x] | [xxx-xxx] | [xx.x-xxx] | |
| Grade 1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | |
| Grade 2 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | |
| Grade 3 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | |
| Fatigue | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxx] | [x:xx-x:xx] | [xxx-xxx] | |
| Total | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | |
| Grade 1 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | |
| Grade 2 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [xxx-xxxx] | [xxx-xxx] | [xxx-xxxx] | |
| Grade 3 | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | |
| | [] | [ ] | [ * * * * * * ] | |

N: total number of subjects in each group; n = Number of subjects; % = Percentage; CI = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabics with anti-malarials to clear parasites; Group 5: Rabics with anti-malarials to prevent infection (prophylaxis).

Solicited AE sac collected on administration and for six days following each injection (Day 1-7).

Denominator for percentage is subjects in safety population.

All confidence intervals are two-sided 95% via Clopper-Pearson method.

Headache, ect.) (Repeat for Fever,

## Protocol No. CVIA-078; RTS,S/AS01 E STATISTICAL ANALYSIS PLAN

Systemic Solicited Adverse Events include: Fever; Headache; Gastrointestinal symptoms (nausea, vomiting, diarrhea and/or abdominal pain); Fatigue; Muscle ache. Each event has intensity scores 0-3 with 0 for no adverse event and 3 for the adverse event that prevents normal activity. For fever, Grade 0: <37.5°C (99.5°F); Grade 1: 37.5°C (99.5°F) to 38.0°C (100.4°F); Grade 2: >38.0°C (>100.4°F) to 39.0°C (102.1°F) (for additional details see protocol)


| | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total |
|---|---|---|---|---|---|---|
| | (N=) | (N=) | (N=) | (N=) | (N<br>=) | (N=) |
| | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] |
| All Systems | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| | [xx.x-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xx.x-xxx] | [xxx-xxx] |
| System Organ Class 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [xx.x-xxx.x] | [xx.x-xx.x] | [xxx-xxxx] | [xx.x-xx.x] | [xx.x-xx.x] |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [x.x.x-x.xx] | [xx.x-xxx] | [xxx-xxxx] | [xx.x-xx.x] | [xx.x-xxx] |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [xx.x-xxx.x] | [xx.x-xx.x] | [xxx-xxxx] | [xx.x-xx.x] | [xx.x-xx.x] |
| Preferred Term 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxx] |
| System Organ Class 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxxx] | [x:xx-x:xx] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] |
| Preferred Term 1 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xx.x-xxx] | [xxx-xxxx] | [xxx-xxx] | [xx.x-xx.x] |
| Preferred Term 2 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xx.x-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] | [xx.x-xx.x] | [xx.x-xx.x] |
| Preferred Term 3 | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [ v v v - v v ] | [v v-v v] | [ * * * * * ] | [ * * * * * * ] | [ * * * * * * ] | [ ^ ^ ^ ^ ^ ] |

(Repeat similarly for other SOCs and PTs)

N: total number of subjects in each group; n = Number of subjects; % = Percentage; CI = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

Subjects who experience one or more episodes of the same adverse event are counted once
All confidence intervals are two-sided 95% via Clopper-Pearson method.

| | (N=)<br>(N=)<br>(N=) | Group 2<br>(N=)<br>n (%) [CI] | Group 3<br>(N=)<br>n (%) [CI] | Group 4<br>(N=)<br>n (%) [CI] | Group 5<br>(N=)<br>n (%) [CI] | Total<br> (N=)<br> n (%) CI |
|---|---|---|---|---|---|---|
| Number of Unsolicited Adverse Events | XXX | XXX | XXX | xxx | xxx | xxx |
| Number of Subjects with any Unsolicited Adverse Events | xx (xx.x%) | (%X.X.X) XX (XX.X/0) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%)<br>[xx.x-xx.x] | (%x.xx) xx |
| Number of Related Unsolicited Adverse Events | XXX | xxx | xxx | xxx | xxx | XXX |
| Number of Subjects with any Related Unsolicited Adverse | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Events | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] |
| Number of Adverse Events of Special Interest (AESIs) | XXX | XXX | XXX | XXX | XXX | XXX |
| Number of Subjects with any Adverse Events of Special | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Interest (AESIs)<br>Number of Related Adverse Events of Special Interest | [XX.X-XX.X] | [XX.X-XX.X] | [XX.X-XX.X] | [XX.X-XX.X] | [XX.X-XX.X] | [XX.X-XX.X] |
| Marriage of Melatea Adverse Events of Special Interest | V. | | ***** | | *************************************** | Y. |
| Number of Subjects with any Related Adverse Events of | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Special Interest | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] |
| Number of Serious Adverse Events (SAEs) | XXX | XXX | XXX | XXX | XXX | XXX |
| Number of Subjects with any Serious Adverse Events (SAEs) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx |
| | [xxx-xxx] | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] |
| Number of Related Serious Adverse Events | XXX | XXX | XXX | XXX | XXX | XXX |
| Number of Subjects with any Related Serious Adverse | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Events | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Number of Serious Adverse Events leading to death. | XXX | XXX | XXX | XXX | XXX | XXX |
| Number of Subjects with any Serious Adverse | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| Events leading to death. | [xxx-xxx] | [xxx-xxx] | [xx.x-xxx] | [xx.x-xx.x] | [xxx-xxx] | [xxx-xxxx] |
| Number of Unsolicited Adverse Events leading to subject discontinuation | XXX | XXX | XXX | xxx | xxx | xxx |
| Number of Subjects with any Unsolicited Adverse Events | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |


# Protocol No. CVIA-078; RTS,S/AS01E STATISTICAL ANALYSIS PLAN

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

All confidence intervals are two-sided 95% via Clopper-Pearson method.

Denominator for percentage is subjects in safety population for whom memory aid data was available.


| Type per n (%) | () n (%) | | (S | (N=) | <u>S</u> |
|---|---|---|---|---|---|
| ted ted 2 gue, Headache, atrointestinal Alass I m 1 2 4 4+ m 2 4 4+ m 2 4 4+ m 2 4 4 4 m 2 4 m 3 4 m 2 4 4 m 2 4 m 3 m 3 m 4 m 4 m 6 m 7 m 7 m 7 m 7 m 8 m 7 m 8 m 7 m 8 m 8 | | n (%)<br>[CI] | n (%) | n (%)<br>[CI] | n (%) |
| at for Swelling at SOI) aic Solicited 2 2 2 3 4 for Fatigue, Headache, ache, Gatrointestinal oms) cited Adverse Events 1 Organ Class 1 ferred Term 1 2 4+ ferred Term 2 3 4+ Annean Class 2 4+ | | | | | |
| at for Swelling at SOI) ie Solicited 2 2 3 if for Fatigue, Headache, ache, Gatrointestinal oms) cited Adverse Events 1 Organ Class 1 ferred Term 1 2 4+ ferred Term 2 3 4+ ferred Term 2 3 4+ ferred Term 2 3 4+ ferred Term 2 4 4+ ferred Term 2 4 4 4 4 4 4 4 4 4 4 4 4 4 | XX | × | X | XX | ×× |
| nic Solicited 2 2 3 4 for Fatigue, Headache, ache, Gatrointestinal oms) cited Adverse Events 1 Organ Class 1 ferred Term 1 2 4+ ferred Term 2 3 4+ ferred Term 2 3 4+ ferred Term 2 4 4- ferred Term 3 4 4- ferred Term 2 4 4- ferred Term 3 4 4- ferred Term 3 4 4- ferred Term 5 4 4- ferred Term 6 4 4 4 4 4 4 4 4 4 4 4 4 4 | | × | XX | XX | XX |
| at for Fatigue, Headache, a che, Gatrointestinal oms) cited Adverse Events 1 Organ Class 1 ferred Term 1 3 4+ ferred Term 2 2 4+ ferred Term 2 3 4+ ferred Term 2 3 4+ | | | | | |
| 2 3 at for Fatigue, Headache, ache, Gatrointestinal oms) cited Adverse Events Organ Class 1 ferred Term 1 2 ferred Term 2 3 4+ ferred Term 2 2 A+ ferred Term 2 3 A+ ferred Term 2 3 A+ ferred Term 2 4 A+ ferred Term 2 3 A+ ferred Term 2 3 A+ ferred Term 2 3 A+ | | | | | |
| e 2 e <del>4</del> 2 e <del>4</del> | xx | X | XX | xx | xx |
| 2 8 4 2 8 4 | XX | X | XX | XX | XX |
| 2 K # 2 K # | | | | | |
| 4 3 2 4 3 2 | | | | | |
| 2 x + 2 x + | | | | | |
| 2 x <sup>‡</sup> 2 x <sup>‡</sup> | | | | | |
| e | xx | XX | XX | XX | XX |
| +<br>+<br>+<br>+<br>+<br>+<br>+<br>+ | xx | X | XX | XX | xx |
| 2 8 4 + | xx | X | XX | XX | xx |
| £ <del>4</del> | xx | X | XX | XX | XX |
| ++ | xx | X | XX | XX | XX |
| System Organ Class 2 | XX | XX | XX | xx | XX |
| System Cigan Ciass 2 | | | | | |
| Preferred Term 1 2 xx | xx | XX | XX | XX | xx |
| 3 xx | xx | X | XX | XX | xx |
| 4+ xx | XX | XX | XX | xx | XX |
| Preferred Term 2 xx | xx | X | XX | XX | xx |
| 3 xx | xx | XX | XX | XX | XX |
| 4+ xx | xx | xx | XX | xx | XX |


N: total number of subjects in each group; n = Number of subjects; "> = Number of subjects; n = Number of subjects; n = Number of subjects; w = Percentage; CI = Confidence interval
Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).
Subjects who experience one or more episodes of the same adverse event are counted once
All confidence intervals are two-sided 95% via Clopper-Pearson method.
Only Adverse Events that have count of occurrences greater than or equal to 2 will be included.

| |
|-------------------------------------|
| Version: 4.0<br>Date: Mar 5th, 2023 |

STATISTICAL ANALYSIS PLAN

Protocol No. CVIA-078; RTS,S/AS01  $_{\rm E}$ 

#### STATISTICAL ANALYSIS PLAN Protocol No. CVIA-078; RTS,S/AS01 $_{\rm E}$

| ion) | | | |
|---|---|---|---|
| (Safety Populati | Total<br>(N=)<br>n (%) [CI] | (%x.xx) xx | [xxx-xxx] |
| Administration | Group 5<br>(N=)<br>n (%) [CI] | (%x.xx) xx | [xxx-xxx] |
| Days Post-IP A | Group 4<br>(N=)<br>n (%) [CI] | (x (%x.xx) xx | [xx.x-xx.x] |
| sted beyond 6 | Group 3<br>(N=)<br>n (%) [CI] | (%x.xx) xx | [xx.x-xx.x] |
| ents that Persi | Group 2<br>(N=)<br>n (%) [CI] n | (%x.xx) xx | [xxx-xxx] |
| ımary of Adverse Ev | Group 1<br>(N=)<br>n (%) CI | (%x.x%) | [xx.x-xx.x] |
| Table 10.4.1.12: Sum | $\begin{array}{cccccccccccccccccccccccccccccccccccc$ | Any Events | |

Total Grade 1 Grade 2 Grade 3

Local

Pain at SOI Total Grade 1

Grade 2 Grade 3

(Repeat for Swelling at SOI)

Systemic

Fever

Total Grade 1 Grade 2 Grade 3

(Repeat for Fatigue, Headache, Muscle ache and gastrointestinal

symptoms)

N: total number of subjects in each group; n = Number of subjects; % = Percentage; CI = Confidence interval

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to clear parasites; Group 6: Rabies with anti-malarials to clear parasites; Group 7: Rabies with anti-malarials with a clear parasites; Group 7: Rabies with a clear parasites; Group 7: Rabies with a clear parasites; Group 7: Rabies with a clear parasites; Group 7: Rabies with a clear parasites; Group 7: Rabies with a clear parasites; Group 7:

Subjects who experience one or more episodes of the same adverse event are counted once

All confidence intervals are two-sided 95% via Clopper-Pearson method.

All solicited Adverse Events that persisted beyond 6 days post-IP administration.


#### STATISTICAL ANALYSIS PLAN Protocol No. CVIA-078; RTS,S/AS01 $_{\rm E}$

| | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total | |
|---|---|---|---|---|---|---|---|
| | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | (N=)<br>n (%) [CI] | P-value |
| Pain at SOI | | | | | | | |
| Yes | x (xx.x%) [xx.x-xxx] | -x.xx] (%x.xx) xx | xx (xx.x%) [xx.x- | | xx (xx.x%) [xx.x | -x.xx] (%x.xx) xx - | 0.xxx |
| No | x (xx.x, xx.x) xx.x [x.xx] | -xxx (xxxx/0%) [xxxx- | xx (xx.x%) [xx.x-<br>xx.x] | x.xx] (%x.xx) xx<br>[x.xx] | xx (xx.x%) [xx.x<br>xx.x] | . xx (xx.x%) [xx.x-<br>xx.x] | |
| Swell at SOI | | | | | | | |
| Yes | x (xx.x%) [xx.x-<br>xx.x] | xx (xx.x%) [xx.x-<br>xx.x] | xx (xx.x%) [xx.x-<br>xx.x] | x (xx.x%) [xx.x-xx xx xx.x] | xx (xx.x%) [xx.x-<br>xx.x] | xx (xx.x%) [xx.x-<br>xx.x] | 0.xxx |
| No | x (xx.x%) [xx.x-xxx] | xx (xx.x%) [xx.x-x-x-x-x-x-x-x-x-x-x-x-x-x-x-x-x-x- | xx (xx.x%) [xx.x- | x (xx.x%) [xx.x-xx] | × | xx (x | |

(Repeat for Fever, Headache, Gastrointestinal symptoms (nausea, vomiting, diarrhea and/or abdominal pain), Fatigue and Muscle ache)

Subjects who experience one or more episodes of the same adverse event are counted once
All confidence intervals are two-sided 95% via Clopper-Pearson method.

p-values are calculated using Fisher's Exact Test.

This table can be expanded to cover other group comparisons, including each preferred terms, grade 4 solicited and unsolicited reactions ect.


| Table 10.4.1.14 | Table 10.4.1.14: Safety Lab Data out of Range (Safety Population) | of Range (Saf | ety Population | | | |
|---|---|---|---|---|---|---|
| | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total |
| | (N=) | (N=) | (N=) | (N=) | (N = 1) | (N |
| | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] |
| Hemoglobin | | | | | | |
| Screening | | | | | | |
| Low | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Normal | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| High | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xx.x-x.x] | [xx.x-x.x] | [xxx-xxx] | [xxx-xxx] |
| Visit 5 | | | | | | |
| Low | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Normal | (%x.xx) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xx.x-xxx] |
| High | (%x.xx) xx | xx (xx.x%) | (%x.xx) xx | (%x.xx) xx | (%x.xx) xx | xx (xx.x%) |
| | [xxx-xxx] | [xx.x-xx.x] | [x.x-x.xx] [x.x-x.xx] [x.x-x.xx] [x.x-x.xx] [x.x-x.xx] | [xx.x-xxx] | [xx.x-xxx] | [xxx-xxx] |

(Repeat for WBC, Platelets, ALT, Creatinine)

N = total number of subjects; %—Percentage; CI = Confidence interval.

N = total number of subjects in each group; n = Number of subjects; %—Percentage; CI = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

All confidence intervals are two-sided 95% via Clopper-Pearson method.


| Table 10.4.1.15: Summary of Safety Lab Kesults (Safety Population) | y Lab Kesuits ( | Satety Populat | 10n) | | | |
|---|---|---|---|---|---|---|
| | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total |
| | (N=) | (N = | (N=) | (N=) | (N=) | (N=) |
| Hemoglobin at Screening | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | [xxx-xxx] | [xxx-xxx] | [xx.x-xxx] | [xx.x-xx.x] | [xxx-xxx] | [xxx-xxx] |
| 95% CI | [xxx-xxx] | | | | [xxx-xxx] | [xxx-xxx] |
| Hemoglobin at Visit 5 | | | | | | |
| n | XX | XX | XX | XX | XX | XX |
| Mean (SD) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xx.x-xx.x] | [xxx-xxx] | [xxx-xxx] |
| 95% CI | [x.x.x-xx.x] | [xxx-xxxx] | [xxx-xxxx] | [xxx-xxx] | [xxx-xxx] | [x.x.x-xx.x] |
| (Compared for WIDC Distalet ALT Compared) | | | | | | |

(Repeat for WBC, Platelet, ALT, Creatinine)

N = total number of subjects in each group.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).

All confidence intervals are two-sided 95% via t-distribution.


| Table 10.4 | Table 10.4.1.16: Summary of Hemoglobinopathy Results (Safety Population) | y of Hemoglob | oinopathy Resu | ilts (Safety Pop | ulation) | |
|---|---|---|---|---|---|---|
| | Group 1 | Group 2 | Group 3 | Group 4 | Group 5 | Total |
| | (N=) | (N=) | (N=) | (N=) | (N=) | (N=) |
| | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] | n (%) [CI] |
| Sickle cell screen | | | | | | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Heterozygous | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| | [xxx-xxx] | [xx.x-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Homozygous | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| G6PD | | | | | | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| | [xxx-xxx] | [xx.x-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Deficient | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | (%x.xx) xx |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Alpha- | | | | | | |
| thalassemia | | | | | | |
| Normal | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Heterozygous | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [xxx-xxx] | [xx.x-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] | [xxx-xxx] |
| Homozygous | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) | xx (xx.x%) |
| | [x.x-x.x] | [xxx-xxx] | [xx-xxx] | [xxx-xxx] | [x.x-x.x] | [xxx-xxx] |

N = total number of subjects in each group; n = Number of subjects; %=Percentage; CI = Confidence interval.
Group 1: RTS,SASOIE with anti-malarials to clear parasites; Group 2: RTS,SASOIE with anti-malarials to clear parasites; Group 4: Rabies with anti-malarials to clear parasites; Group 4: Rabies with anti-malarials to clear parasites; Group 5: Rabies with anti-malarials to prevent infection (prophylaxis).
All confidence intervals are two-sided 95% via Clopper-Pearson method.


| | ı |
|---|---|
| | ı |
| | ı |
| | ı |
| | ı |
| | ı |
| ! | ı |
| ! | ı |
| i | ı |
| ! | ı |
| 1 | ı |
| | ı |
| | ı |
| | ı |
| | ı |
| | ı |
| | ı |
| | ı |
| 1 | ı |
| | ı |
| 1 | ı |
| 1 | ı |
| | ı |
| | ı |
| | ı |
| | ı |
| | ı |
| ) | |

Total (N=) n (%) [CI]

Group 5 (N=) n (%) [CI]

| reening | | | | | | |
|----------|---|---|---|---|---|---|
| Positve | × | × | × | × | × | × |
| Negative | × | × | × | × | × | × |
| N/A | × | × | × | × | × | × |
| sit 2 | | | | | | |
| Positve | × | × | × | × | × | × |
| Negative | × | × | × | × | × | × |
| N/A | × | × | × | × | × | × |
| Visit 5 | | | | | | |
| Positve | × | × | × | × | × | × |
| Negative | × | × | × | × | × | × |
| N/A | × | × | × | × | × | × |

Repeat for Visit 8

N = total number of subjects in each group; n = Number of subjects; %=Percentage; CI = Confidence interval.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabics with anti-malarials to clear parasites; Group 5: Rabics with anti-malarials to clear parasites; Group 7: Rabics with anti-malarials to clear parasites.


#### STATISTICAL ANALYSIS PLAN Protocol No. CVIA-078; RTS,S/AS01 $_{\rm E}$

| | 1 | | ı | i | |
|---|---|---|---|---|---|
| | Total | (N=) | n (%) [CI] | (%x.xx) xx | [x.x-x.x] |
| ty Population) | Group 5 | (N=) | n (%) [CI] | ( (%x.xx) xx | [xxx-xxx] |
| eatment (Safe | Group 4 | (N=) | n (%) [CI] | x (%x.xx) xx | [xxx-xxx] |
| e Events by Tr | Group 3 | (N=) | n (%) [CI] | x (%x.xx) xx | [xxx-xxx] |
| erious Advers | Group 2 | (N=) | n (%) [CI] | (%x.xx) xx | [xxx-xxx] |
| nary of All Non-S | Group 1 | (N=) | n (%) [CI] | (%x.xx) xx | [xxx-xxx] |
| Table 10.4.1.18: Summary of All Non-Serious Adverse Events by Treatment (Safety Population) | | | | All Non-Serious Adverse | Events |

Preferred Term 2 Preferred Term 3 Preferred Term 1

System Organ Class 1

System Organ Class 2

Preferred Term 1 Preferred Term 2

Preferred Term 3

 $N = total\ number\ of\ subjects;\ \% = Percentage;\ CI = Confidence\ interval.$ 

Denominator for percentage is subjects in the safety population.

Subjects who experience one or more episodes of the same adverse event are counted once.

Solicited AEs are included in the table within categories of system organ class and preferred term.

All confidence intervals are two-sided 95% via Clopper-Pearson method.

Group 1: RTS,S/AS01E with anti-malarials to clear parasites; Group 2: RTS,S/AS01E with anti-malarials to prevent infection (prophylaxis); Group 3: RTS,S/AS01E without anti-malarials to clear parasites; Group 5: Rabics with anti-malarials to clear parasites; Group 5: Rabics with anti-malarials to clear parasites; Group 6: Rabics with anti-malarials to clear parasites; Group 7: Rabics with anti-malarial to clear parasites; Group 7: Rabics with anti-malarial to clear parasites; Group 7: Rabics with anti-malarial to clear parasites; Group 7: Rabics with anti-malarial to clear parasi


### STATISTICAL ANALYSIS PLAN

#### 12. DEMOGRAPHICS LISTINGS

Listing 10.1.1: Protocol Deviations

| trief Description | |
|-------------------|------------|
| I I | XXXXXXXXX |
| Category | XXXX |
| Date Reported | ddMMMyyyy |
| Date Occurred | ddMMMyyyy |
| Group | Groups 1-5 |
| Subject ID | XXXXX |

The following deviation categories are included for the study:
Eligibility
Informed consent
Randomization error
Antimalarial drugs administered incorrectly
IP administered incorrectly
IP administration missed

Missed visit
Out-of-window visit
Specimen not collected
Procedure done incorrectly
Procedure not done
Other


## Protocol No. CVIA-078; RTS,S/AS01<sub>E</sub> STATISTICAL ANALYSIS PLAN

| Listi | ng 10.1.2: Enrol | ment Statu | ıs, Demographic | s and Subj | ect Disposition | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Informed | | | | | | | | | |
| | Consent Signed | | | | | | | | Date of | |
| | Date of | | | | | | | | Completion/ | |
| | Informed | | | | Reactogenicity | | | Completed | Early | |
| Subject ID | Subject ID Consent E | | ligible Randomized Group | Group | Cohorts? | Sex/Age (Years) | Race/Ethnicity | | Termination | |
| XXX | Yes/xxxxx | No | No | XXX | (Yes/No) | Female/39 | xxx/xxx | No | xxxx | XXXXXXXXXXXXX |
| XXX | xxx Yes/xxxxxx | Yes | Yes | XXX | | XXX | XXX/XXX | Yes | XXXX | |


| STATISTICAL ANALYSIS PLAN |
|-------------------------------------|
| Protocol No. CVIA-078; RTS,S/AS01 E |

Listing 10.1.3: Eligibility Criteria Not Met

| | dy protocol from if study vaccine. | |
|---|---|---|
| Criteria Description Subject has provided signed or thumb printed and dated informed consent form. XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Subject has planned administration/administration of a vaccine not foreseen by the study protocol from within 30 days before the first dose of study vaccine until 30 days after the last dose of study vaccine. XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Confidential |
| Eligibility Criteria<br>Inclusion Criteria | Exclusion Criteria | Version: 4.0 Date: Mar 5th 2023 |
| Subject ID<br>xxxxx | | Version: 4.0 |

### Protocol No. CVIA-078; RTS,S/AS01 E STATISTICAL ANALYSIS PLAN

| Criteria |
|-------------|
| Eligibility |
| g of All |
| : Listing |
| g 10.1.4 |
| Listing |

| Спепа Бееприон | Subject has provided signed or thumb printed and dated informed consent form. | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Subject has planned administration/administration of a vaccine not foreseen by the study protocol from within 30 days before the first dose of study vaccine until 30 days after the last dose of study vaccine. XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
|---|---|---|---|
| Engionny Criteria | Inclusion Criteria | | Exclusion Criteria |


| STATISTICAL ANALYSIS PLAN |
|-------------------------------------|
| Protocol No. CVIA-078; RTS,S/AS01 E |

| | | BMI (unit) | ×××× |
|---|---|---|---|
| | Weight | (unit) Height (unit) BMI (unit) | x.xx.x |
| | | (unit) | XXX |
| | | Sex Ethnicity | XXXXXX |
| | | Sex | × |
| graphics | | Race | XXXXXX |
| Listing 10.1.5: Baseline Demographics | | Age (years) | × |
| ; 10.1.5: 1 | | Group | XX |
| Listing | | Subject ID Group Age (years) Race | XXXXX |


| | TICAL ANALYSIS |
|---|-----------------|
| | STAT |
| | A-078; RTS,S/AS |
| , | otocol No. |

| | HLA Typing | Date/Time | HLA-A |
|---|---|---|---|
| Listing 10.1.6: HIV Status and HLA Typing | Buccal Swab | Date/Time | ddMMMyyyy/hh:mm |
| | HIV Test | HIV Status | Negative/Positive |
| | | Subject ID Group Date/Time | xxx ddMMMyyyy/hh:mm Negative/Positive ddMMMyyyy/hh:mm HLA-A |
| | | Group | XXX |
| Listin | | Subject ID | xxxxx |


| | Route/ Freq | xxxx/xxxx |
|---|---|---|
| | Dose/ Unit | xxx/xxx |
| | Start Date/ End ATC Level 4/ Preferred Date Term/ Medication Name | xxx/xxx/xxxx |
| Listing 10.1.7: Prior Medications | Start Date/ End<br>Date | xxxx ddMMMyyyy/<br>(ddMMMyyyy) |
| ng 10.1.7: ] | Group | XXXX |
| Listi | Subject ID Group | Xxx |


| | | Route/ Freq | | | xxxx/xxxx |
|---|---|---|---|---|---|
| | | Dose/ Unit | | | xxx/xxxx |
| | ATC Level 4/ Preferred | Term/ Medication Name | | | xxx/xxx/xxx |
| isting 10.1.8: Concomitant Medication | Start Date/ End A | Date | ddmmmyyyy/ | (ddmmmyyyy or | ONGOING) |
| 0.1.8: Concomit | | Group | | | XXXX |
| Listing 1 | | Subject ID | | | Xxx |


| List | ing 10.1.9: | Listing 10.1.9: Medical History | | |
|---|---|---|---|---|
| | Group | Start Date / End | | |
| Subject ID | | Date | System Organ Class | Preferred Term |
| | | ddMMMyyyy / | | |
| | | ddMMMyyyy or | | |
| Xxxx | XXXX | ongoing | XXXXXX | XXXXXXX |
| | | ddMMMyyyy / | | |
| | | ddMMMyyyy or | | |
| | | ongoing | | |

 Version: 4.0 Date: Mar 5th, 2023 Repeat until Visit 18

Visit 9

Visit 8

 (Yes/No)
 (Yes/No)
 (Yes/No)
 (Yes/No)
 (Yes/No)

Treatment and immunization (Epoch 1)

Visit 6

Visit 5

Visit 4

Visit 3

Subject ID Group

(Yes/No) Visit 2

XXXX

XXXX

Listing 10.1.10.1: Visit Attendance (Epoch 1)

| oĮ |
|------|
| 95 |
| Page |


| Active Detection of Infection (Epoch 2) | Active Detection of Infection (Epoch 2) |
| Visit 19 | Visit 21 | Visit 22 | Visit 24 | Visit 25 | Visit 27 |
| (Yes/No)

Listing 10.1.10.2: Visit Attendance (Epoch 2)

Group

Subject ID

| Version: 4.0 | Confidential |
|---------------------|--------------|
| Date: Mar 5th, 2023 | |

| (Epoch 3) |
|-------------------------|
| Infection-Extension (Ep |

| | | Visit 35 | (Yes/ No) |
|------------------|------------------|----------------------------|-----------|
| | 13) | Visit34 | (Yes/ No) |
| | ension (Epoch 3) | Visit 33 | (Yes/ No) |
| | Infection-Ext | Visit 30 Visit 31 Visit 32 | (Yes/ No) |
| | e Detection of | Visit 31 | (Yes/ No) |
| | Activ | Visit 30 | (Yes/No) |
| (Epoch 3) | | Visit 29 | (Yes/No) |
| Visit Attendance | | Visit 28 V | (Yes/No) |
| ng 10.1.10.3: | C. 2011 | dinois | XXXX |
| Listi | Cubicot ID | an palanc | XXXX |


Listing 10.1.11: Vaccine administration

| 1 | |
|------------------|-----------|
| Vaccination Date | ddMMMyyyy |
| Vaccine Dose | xxx |
| Visit Number | Xxx |
| Group | XXXX |
| Subject ID | XXXX |


| | Full dose? | | (Yes/No) |
|-------------------|-------------------|------------------|-----------------|
| | Number of | tablets returned | x |
| | Number of tablets | dispensed | × |
| | | Date/Time | ddMMMyyyy;hh:mm |
| | Anti-Malarials | Taken | XXX |
| 2: Anti-Malarials | | Visit Number | Xxx |
| ng 10.1.12: | | Group | XXXX |
| Listi | | Subject ID | XXXX |


| Group Parameter Visit Date: Time Screening Screening ddmnmyyyy; hh:mm Visit 5 ddmnmyyyy; hh:mm Visit 11 ddmnmyyyy; hh:mm Visit 11 ddmnmyyyy; hh:mm Visit 17 ddmnmyyyy; hh:mm Blood Screening Pressure (Visit 1 or 2) Visit 5 ddmmmyyyy; hh:mm Visit 6 ddmmmyyyy; hh:mm | Results (Units) |
|---|---|
| Screening Pulse Rate (Visit 1 or 2) Visit 5 Visit 8 Visit 11 Visit 11 Visit 17 Systolic Screening Pressure (Visit 1 or 2) | |
| Pulse Rate (Visit 1 or 2) Visit 5 Visit 8 Visit 11 Visit 17 Systolic Blood Screening Pressure (Visit 1 or 2) | |
| Visit 5 Visit 8 Visit 11 Visit 17 Screening (Visit 1 or 2) Visit 5 | |
| Visit 8 Visit 11 Visit 17 Screening (Visit 1 or 2) | |
| Visit 11 Visit 17 Screening (Visit 1 or 2) | |
| Visit 17 Screening (Visit 1 or 2) Visit 5 | |
| Screening (Visit 1 or 2) Visit 5 | n |
| Screening (Visit 1 or 2) | п |
| Screening (Visit 1 or 2) Visit 5 | |
| (Visit 1 or 2)<br>Visit 5 | |
| | (mmHg)) |
| | n xxx (mmHg)) |
| Visit 8 ddmmmyyyy: hh:mm | n xxx (mmHg)) |
| | n xxx (mmHg)) |
| Visit 17 ddmmmyyyy: hh:mm | n xxx (mmHg)) |

| for | _ | 9 |
|----------|-------|--------|
| Repeat f | other | peidus |


### Protocol No. CVIA-078; RTS,S/AS01E STAT

1<sub>E</sub> STATISTICAL ANALYSIS PLAN

#### Listing 10.1.14: Physical Examinations

| | | | | | Results/ | Clinically |
|---|---|---|---|---|---|---|
| Subject ID | Group | Group Body System | Visit | Date/Time of Exam | Description | Significant? |
| XXXXX | Х | Abdomen | Screening | ddmmmyyyy:hh:mm | Normal | (Yes/No) |
| | | | Visit 5 | ddmmmyyyy;hh:mm | Normal | (Yes/No) |
| | | | Visit 11 | ddmmmyyyy;hh:mm | Normal | (Yes/No) |
| | | | | ddmmmyyyy:hh:mm | | (Yes/No) |
| | | Repeat other body systems | | | | |

Repeat other subjects


13. SAFETY LISTINGS
Listing 10.2.1: Solicited Adverse Events (Safety Population)

| Days from Most<br>Recent | * Vaccination** | 2 | 33 | 1 |
|---|---|---|---|---|
| Duration | (in days) * | xxxx | XXXX | XXXX |
| | Stop Date | | XXXX | XXXX |
| | Start Date | xxx | XXX | XXX |
| | Maximum Severity Start Date | Grade 2 | Grade 1 | Grade 1 |
| | AE Term | Pain at SOI | Swelling at SOI | Headache |
| | Type | Local | | Systemic |
| Reported at | Visit | xxx | | |
| | Group | | | |
| | Subject ID Group | XXXXX | | |


<sup>\*</sup> Duration= AE stop date – AE start date + 1 \*\* Difference between AE start date and most recent vaccination date + 1.


Listing 10.2.2: Unsolicited Adverse Events (Safety Population)

| | | SAE? | |
|---|---|---|---|
| | | AESI? | |
| Action Taken with<br>Study<br>Treatment/Action | y Taken with | Antimalarials | |
| Severity/ | nt Relation to Study | Treatment | |
| | Days from Most Recent Relation to Study | Vaccination** Treatment Antimalarials AESI? SAE? | |
| | Duration | (in days) * | |
| | Outcome/ | Outcome Date | |
| | Start | Date | |
| | System Organ | Class Date ( | |
| | | AE Term | XXX |
| | | Group | XXX |
| | Subject | ID Group AE Ter | XXXXX |


Listing 10.2.3: Serious Adverse Events (Safety Population)

| | | se | 'n | |
|---|---|---|---|---|
| | | Serious Advers | Event Categor | |
| | | Action Taken with | Study Treatment? | |
| | Severity/ | Relation to Study | Treatment | |
| | | Days from Most | Recent Vaccination** | |
| | | Duration | (in days) * | |
| | | Outcome/ | Outcome Date | |
| = | | Start | Date | |
| MedDRA Preferre | Term/ | System Organ | Class | |
| | | ΑE | Term | XXX |
| | | | Group | XXX |
| | | Subject | Π | XXXXX |

| | | Serious Adverse | Event? | |
|---|---|---|---|---|
| | | Action Taken with | Study Treatment? | |
| | Severity/ | Relation to Study | Treatment | |
| | | Duration Days from Most Relation to Study Action Taken with Serious Adverse | ID Group Term Class Date Outcome Date (in days)* Recent Vaccination** Treatment Study Treatment? Event? | |
| ation) | | Duration | (in days) * | |
| erest (Safety Popul | | Outcome/ | Outcome Date | |
| ecial Int | _ | Start | Date | |
| isting 10.2.4; Adverse Events of Special Interest (Safety Population) | MedDRA Preferred<br>Term/ | System Organ | Class | |
| 0.2.4: AG | | ΑE | Term | XXX |
| Listing 1 | | | Group | XXX XXX |
| | | Subject | П | XXXXX |

\* Duration= AE stop date – AE start date + 1 \*\* Difference between AE start date and most recent vaccination date + 1.


| | Normal/<br>Abnormal | Normal | Normal |
|------------------|---------------------|------------|------------|
| ou) | Results | XX | XX |
| (Safety Populati | Date | ddMMMyyyy | ddMMMyyyy |
| Results | Visit | 1 | 2 |
| ty Laboratory | Test Name | Hemoglobin | Hemoglobin |
| .5: Safe | Sex | XXX | XXX |
| sting 10.2 | Group | XXX | XXX |
| Ξ | Subject ID | XXXXX | XXXXX |


Listing 10.2.6: Hemoglobinopathy Tests Results (Safety Population)

Results

Date
ddMMMyyyy
ddMMMyyyy

 Subject ID
 Group
 Sex
 Test Name

 xxxxx
 xxx
 Sickle Cell Screen

 xxx
 xxx
 G6P

 xxx
 xxx
 Apha-thalassemia

Repeat for other subjects


Listing 10.2.7: Urine Pregnancy Tests for Female Subjects (Safety Population)

Results
Negative
Negative
Negative
Negative
Negative

Date
ddMMMyyyy
ddMMMyyyy
ddMMMyyyy
ddMMMyyyy

X X X

Repeat for other subjects

Group

XXX XXX

| ıtial |
|-----------|
| nfidentia |
| Con |
Protocol No. CVIA-078; RTS,S/AS01  $_{\rm E}$ 

STATISTICAL ANALYSIS PLAN

### 15. VACCINE EFFICACY LISTING Listing 10.4.1 Listing of First Infection Events (FIEs)

| Event | Yes/No |
|------------------------------------------------------------|-----------|
| At Risk Time<br>(yrs) | X.XX |
| End Date at Risk | ddMMyyyy |
| Start Date at Risk End Date at Risk At Risk Time (yrs) | ddMMMyyyy |
| Per Protocol<br>Population for<br>Efficacy | Y. |
| Group | Group 1 |
| Subject ID | XXXXX |


# Protocol No. CVIA-078; RTS,S/AS01<sub>E</sub> STATISTICAL ANALYSIS PLAN

Listing 10.4.2 Listing of Parasitemia Test Results (ADI)

| Subject ID | Group | Visit | Date of Sample<br>Collection | Parasitemia Test Results |
|---|---|---|---|---|
| XXXXX | Group 1 | Visit 19 | ddMMMyyyy | Positive/Negative |


| | |
|---|---|
| 16. DEMOGRAPHICS FIGURES Figure 10.1.1: CONSORT Diagram | Version: 4.0<br>Date: Mar 5th, 2023 |

STATISTICAL ANALYSIS PLAN

Protocol No. CVIA-078; RTS,S/AS01  $\rm _E$ 

## CONSORT Diagram for CVIA 078 RTS, S/AS01<sub>E</sub>




### 17. VACCINE EFFICACY FIGURES

Figure 10.2.1: Kaplan-Meier survival curve for FIEs in Groups 1 and 4.




STATISTICAL ANALYSIS PLAN

Figure 10.2.2: Kaplan-Meier survival curve for FIEs in Groups 1 and 4 stratified by HIV status.





Figure 10.2.3: Kaplan-Meier survival curve for FIEs in Groups 2 and 5.




STATISTICAL ANALYSIS PLAN

Figure 10.2.4: Kaplan-Meier survival curve for FIEs in Groups 2 and 5 stratified by HIV status.



Repeat the same survival curves for groups 1 and 2, groups 4 and 5

Figure 10.2.5: Kaplan-Meier survival curve for FIEs in Groups 1 and 2 Figure 10.2.6: Kaplan-Meier survival curve for FIEs in Groups 4 and 5 Confidential Date: Mar 5th, 2023 Version: 4.0


STATISTICAL ANALYSIS PLAN

Figure 10.2.7: Scaled Schoenfeld residuals with 95% confidence interval versus time for Groups 1 and 4 FIEs during the entire study period (ATP cohort for efficacy)



p-value=x.xxx


Date: Mar 5th, 2023


Figure 10.2.8: Scaled Schoenfeld residuals with 95% confidence interval versus time for Groups 2 and 5 FIEs during the entire study period (ATP cohort for efficacy)



p-value=x.xxx

Repeat the same residual plots for groups 1 and 2, groups 4 and 5:

Figure 10.2.9: Scaled Schoenfeld residuals with 95% confidence interval versus time for Groups 1 and 2 FIEs during the entire study period (ATP cohort for efficacy)
Figure 10.2.10: Scaled Schoenfeld residuals with 95% confidence interval versus time for Groups 4 and 5 FIEs during the entire study period (ATP cohort for efficacy).

Confidential Version: 4.0


## SO1E STATISTICAL ANALYSIS PLAN

#### 18. IMMUNOGENICITY FIGURES

Figure 10.3.1: Reverse Cumulative Distribution Curves for Anti-CS NANP Antibody Titers in Each Group (ATP cohort for immunogenicity)

F10.2.5 Reverse Cumulative Distribution Curve for Anti-CS NANP Antibody Titers Efficacy Population for Immunogenicity



Repeat the same plots for Anti-CS C-terminal and Anti-HBsAb titers in Figures 10.2.6 and 10.2.7

Figure 10.3.2: Reverse Cumulative Distribution Curves for Anti-CS C-term Antibody Titers in Each Group (ATP cohort for immunogenicity)
Figure 10.3.3: Reverse Cumulative Distribution Curves for Anti-HBsAb Titers in Each Group (ATP cohort for immunogenicity)

Confidential Version: 4.0

Date: Mar 5th, 2023

